CLINICAL TRIAL: NCT02315703
Title: A Phase 1/2a Trial to Evaluate the Safety/Tolerability and Immunogenicity of Homologous Ad26 Mosaic Vector Regimens or Ad26 Mosaic and MVA Mosaic Heterologous Vector Regimens, With High-Dose, Low-Dose or no Clade C gp140 Protein Plus Adjuvant for HIV Prevention
Brief Title: Safety, Tolerability, and Immunogenicity Study of Homologous Ad26 Mosaic Vector Vaccine Regimens or Heterologous Ad26 Mosaic and MVA Mosaic Vector Vaccine Regimens With Glycoprotein 140 (gp140) for Human Immunodeficiency Virus (HIV) Prevention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); US Military HIV Research Program (Network); Beth Israel Deaconess Medical Center (Other); International AIDS Vaccine Initiative (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR106152; HIV-V-A004 (Other: Janssen Vaccines & Prevention B.V.); IPCAVD009 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; Acquired Immuno-Deficiency Syndrome; Acquired Immunodeficiency Syndrome Virus; adenovirus serotype 26; Ad26.Mos.HIV; Modified Vaccinia Ankara; Glycoprotein; Adjuvant; Vaccine; Placebo
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group 1 (Experimental): Participants will receive adenovirus serotype 26-Mosaic -Human Immunodeficiency Virus (Ad26.Mos.HIV) vaccine at Week 0 and 12; followed by Ad26.Mos.HIV vaccine + HIV type 1 Clade C glycoprotein 140 drug product (gp140 DP) vaccine containing 250 microgram (mcg) of total protein mixed with adjuvant (aluminum phosphate) at Week 24 and 48.
  Interventions: Biological: Ad26.Mos.HIV; Biological: gp140 DP High-dose
- Group 2 (Experimental): Participants will receive Ad26.Mos.HIV vaccine at Week 0 and 12; followed by Ad26.Mos.HIV vaccine + gp140 DP vaccine containing 50 mcg of total protein mixed with adjuvant at Week 24 and 48.
  Interventions: Biological: Ad26.Mos.HIV; Biological: gp140 DP Low-dose
- Group 3 (Experimental): Participants will receive Ad26.Mos.HIV vaccine at Week 0 and 12; followed by Ad26.Mos.HIV vaccine + placebo injection at Week 24 and 48.
  Interventions: Biological: Ad26.Mos.HIV; Drug: Placebo
- Group 4 (Experimental): Participants will receive Ad26.Mos.HIV vaccine at Week 0 and 12; followed by modified Vaccinia Ankara (MVA)-Mosaic vaccine + gp140 DP vaccine containing 250 mcg of total protein mixed with adjuvant at Week 24 and 48.
  Interventions: Biological: Ad26.Mos.HIV; Biological: MVA-Mosaic; Biological: gp140 DP High-dose
- Group 5 (Experimental): Participants will receive Ad26.Mos.HIV vaccine at Week 0 and 12; followed by MVA-Mosaic vaccine + gp140 DP vaccine containing 50 mcg of total protein mixed with adjuvant at Week 24 and 48.
  Interventions: Biological: Ad26.Mos.HIV; Biological: MVA-Mosaic; Biological: gp140 DP Low-dose
- Group 6 (Experimental): Participants will receive Ad26.Mos.HIV vaccine at Week 0 and 12; followed by MVA-Mosaic vaccine + placebo injection at Week 24 and 48.
  Interventions: Biological: Ad26.Mos.HIV; Biological: MVA-Mosaic; Drug: Placebo
- Group 7 (Experimental): Participants will receive Ad26.Mos.HIV vaccine at Week 0 and 12; followed by gp140 DP vaccine containing 250 mcg of total protein mixed with adjuvant + placebo injection at Week 24 and 48.
  Interventions: Biological: Ad26.Mos.HIV; Biological: gp140 DP High-dose; Drug: Placebo
- Group 8 (Placebo Comparator): Participants will receive 1 placebo injection at Week 0 and 12; followed by 2 placebo injections at Week 24 and 48.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ad26.Mos.HIV — Recombinant replication-deficient Ad26 vectored vaccine and consists of 3 Ad26 vectors, one containing a mosaic insert of envelop (Env) sequence, and 2 vectors containing mosaic inserts of Gag and Pol sequences (Ad26.Mos.1.Env + Ad26.Mos1.Gag-Pol + Ad26.Mos2.Gag-Pol). Total dose is 5*10^10 viral particle per 0.5 milliliter (mL) injection administered intramuscularly.
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5; Group 6; Group 7
Biological: MVA-Mosaic — Recombinant live attenuated MVA virus-vectored vaccine that has been genetically engineered to express 2 mosaic Gag, Pol, and Env sequences (Mosaic 1 and Mosaic 2). Total dose is 10^8 plaque-forming unit per 0.5 mL injection administered intramuscularly.
  Arms: Group 4; Group 5; Group 6
Biological: gp140 DP Low-dose — The gp140 DP vaccine containing 50 mcg of total protein, mixed with aluminum phosphate adjuvant (0.425 mg aluminum), per 0.5 mL injection administered intramuscularly.
  Arms: Group 2; Group 5
Biological: gp140 DP High-dose — The gp140 DP vaccine containing 250 mcg of total protein, mixed with aluminum phosphate adjuvant, per 0.5 mL injection administered intramuscularly.
  Arms: Group 1; Group 4; Group 7
Drug: Placebo — Normal saline, 0.5 mL injection administered intramuscularly.
  Arms: Group 3; Group 6; Group 7; Group 8

SUMMARY:
The purpose of this study is to assess the safety and tolerability of various regimens containing adenovirus serotype 26-Mosaic -Human Immunodeficiency Virus (Ad26.Mos.HIV), Modified Vaccinia Ankara (MVA)-Mosaic, and/or HIV type 1 Clade C glycoprotein 140 drug product (gp140 DP) components and to compare envelope binding antibody responses between the different vaccine regimens.

DETAILED DESCRIPTION:
This is a multicenter (more than 1 hospital or medical school team work on a study), randomized (the study drug is assigned by chance), parallel group (each group of participants will be treated at the same time), placebo-controlled (study in which the experimental treatment or procedure is compared to a pretend treatment with no drug in it to test if the drug has a real effect), and double-blind (neither physician nor participant knows the treatment that the participant receives) study. All eligible participants will be randomly assigned to receive 1 of the 8 vaccine regimens. Participants will receive study vaccines (Ad26.Mos.HIV, MVA-Mosaic, gp140 DP, and placebo) 4 times as per assigned regimen. The study comprises a Screening Period (up to 4 weeks), a Vaccination Period (participants will be vaccinated at Baseline (Week 0), Week 12, Week 24 and Week 48), and a Follow-up Period (up to 48 weeks). A long-term follow-up period (approximately 2 years after Week 96) will continue for participants randomized to the regimen subsequently selected for future studies, based on analysis of Week 28 data. If Week 28 data are inconclusive, Week 52 data will be considered for regimen selection. If no clear decision can be made, the extended follow-up period could include participants from more than 1 group for assessing durability of immune responses. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy on the basis of physical examination, medical history, electrocardiogram (ECG) and laboratory criteria, and vital signs measurement performed at Screening
* Participants are negative for human immunodeficiency virus (HIV) infection at Screening
* All female participants of childbearing potential must have a negative serum (beta human chorionic gonadotropin) at Screening, and a negative urine pregnancy test pre-dose on Week 0, 12, 24, and 48
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction until 3 months after receiving the last dose of study vaccine. A man must agree not to donate sperm until 3 months after receiving the last dose of study vaccine
* Participants are assessed by the clinic staff as being at low risk for HIV infection

Exclusion Criteria:

* Participant has chronic active hepatitis B or active hepatitis C, active syphilis infection, chlamydia, gonorrhea, or trichomonas. Active syphilis documented by exam or serology unless positive serology is due to past treated infection
* In the 12 months prior to enrollment, participant has a history of newly acquired herpes simplex virus type 2 (HSV-2), syphilis, gonorrhea, non-gonococcal urethritis, chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranulomavenereum, chancroid, or hepatitis B
* Participant has any clinically significant acute or chronic medical condition that in the opinion of the investigator would preclude participation (for example, history of seizure disorders, bleeding/clotting disorder, autoimmune disease, active malignancy, poorly controlled asthma, active tuberculosis or other systemic infections)
* Participant has had major surgery within the 4 weeks prior to study entry or planned major surgery through the course of the study
* Participant has had a thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Participant has a history of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow up)
* Participant has an ECG (per examination and interpretation of a cardiologist) with clinically significant findings, or features that would interfere with the assessment of myo/pericarditis, including any of the following: a) conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS >=120 millisecond [ms], PR interval >=220 ms, any 2nd or 3rd degree AV block, or QTc prolongation [>450 ms]); b) significant repolarization (ST segment or T wave) abnormality; c) significant atrial or ventricular arrhythmia, frequent atrial or ventricular ectopy (for example frequent premature atrial contractions, 2 premature ventricular contractions in a row); d) ST elevation consistent with ischemia, or evidence of past or evolving myocardial infarction
* Participant has a history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products, or neomycin or streptomycin or egg products

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 393 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trials, Study Director — Janssen Vaccines & Prevention B.V.
Locations (12):
- United States (5):
  - Aurora, Colorado
  - Miami, Florida
  - Rockville, Maryland
  - Boston, Massachusetts
  - Austin, Texas
- Kigali, Rwanda
- South Africa (3):
  - Cape Town
  - Durban
  - Johannesburg
- Bangkok, Thailand
- Uganda (2):
  - Entebbe
  - Kampala

REFERENCES:
- [Derived] van Duijn J, Stieh D, Fernandez N, King D, Gilmour J, Tolboom J, Callewaert K, Willems W, Pau MG, De Rosa SC, McElrath MJ, Barouch DH, Hayes P. Mosaic HIV-1 vaccination induces anti-viral CD8+ T cell functionality in the phase 1/2a clinical trial APPROACH. J Virol. 2023 Oct 31;97(10):e0112623. doi: 10.1128/jvi.01126-23. Epub 2023 Oct 9. PMID 37811993
- [Derived] Barouch DH, Tomaka FL, Wegmann F, Stieh DJ, Alter G, Robb ML, Michael NL, Peter L, Nkolola JP, Borducchi EN, Chandrashekar A, Jetton D, Stephenson KE, Li W, Korber B, Tomaras GD, Montefiori DC, Gray G, Frahm N, McElrath MJ, Baden L, Johnson J, Hutter J, Swann E, Karita E, Kibuuka H, Mpendo J, Garrett N, Mngadi K, Chinyenze K, Priddy F, Lazarus E, Laher F, Nitayapan S, Pitisuttithum P, Bart S, Campbell T, Feldman R, Lucksinger G, Borremans C, Callewaert K, Roten R, Sadoff J, Scheppler L, Weijtens M, Feddes-de Boer K, van Manen D, Vreugdenhil J, Zahn R, Lavreys L, Nijs S, Tolboom J, Hendriks J, Euler Z, Pau MG, Schuitemaker H. Evaluation of a mosaic HIV-1 vaccine in a multicentre, randomised, double-blind, placebo-controlled, phase 1/2a clinical trial (APPROACH) and in rhesus monkeys (NHP 13-19). Lancet. 2018 Jul 21;392(10143):232-243. doi: 10.1016/S0140-6736(18)31364-3. Epub 2018 Jul 6. PMID 30047376

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Ad26/Ad26 + gp140 High Dose (HD): Participants received 5*10^10 viral particle (vp) of adenovirus serotype 26- Mosaic -Human Immunodeficiency Virus (Ad26.Mos.HIV) Intramuscular (IM) vaccine at Week 0 and 12. At Week 24 and 48, participants received 5*10^10 vp Ad26.Mos.HIV vaccine and HIV type 1 Clade C glycoprotein 140 drug product (gp140 DP) IM high dose vaccine containing 250 microgram (mcg) of total glycoprotein mixed with adjuvant (aluminum phosphate). Participants in Group 1 and 2 who received all 4 vaccinations in main study continued in long-term extension (LTE) phase after Week 96 up to Week 336.
- Group 2: Ad26/Ad26 + gp140 Low Dose (LD): Participants received 5*10^10 vp of Ad26.Mos.HIV IM vaccine at Week 0 and 12. At Week 24 and 48, participants received 5*10^10 vp Ad26.Mos.HIV vaccine and gp140 DP IM low dose vaccine containing 50 mcg of total glycoprotein mixed with adjuvant (aluminum phosphate). Participants in Group 1 and 2 who received all 4 vaccinations in main study continued in long-term extension (LTE) phase after Week 96 up to Week 336.
- Group 3: Ad26/Ad26: Participants received 5*10^10 vp of Ad26.Mos.HIV IM vaccine at Week 0 and 12. At Week 24 and 48, participants received 5*10^10 vp Ad26.Mos.HIV IM vaccine and matched placebo IM vaccine.
- Group 4: Ad26/MVA + gp140 HD: Participants received 5*10^10 vp of Ad26.Mos.HIV IM vaccine at Week 0 and 12. At Week 24 and 48, participants received 10^8 plaque-forming unit (pfu) modified Vaccinia Ankara (MVA)-Mosaic IM vaccine and gp140 DP IM high dose vaccine containing 250 mcg of total glycoprotein mixed with adjuvant.
- Group 5: Ad26/ MVA + gp140 LD: Participants received 5*10^10 vp of Ad26.Mos.HIV IM vaccine at Week 0 and 12. At Week 24 and 48, participants received 10^8 pfu MVA-Mosaic IM vaccine and gp140 DP IM low dose vaccine containing 250 mcg of total glycoprotein mixed with adjuvant.
- Group 6: Ad26/MVA: Participants received 5*10^10 vp of Ad26.Mos.HIV IM vaccine at Week 0 and 12. At Week 24 and 48, participants received 10^8 pfu MVA-Mosaic IM vaccine and matched placebo IM vaccine.
- Group 7: Ad26/ gp140 HD: Participants received 5*10^10 vp of Ad26.Mos.HIV IM vaccine at Week 0 and 12. At Week 24 and 48, participants received gp140 DP IM high dose vaccine containing 250 mcg of total glycoprotein mixed with adjuvant (aluminum phosphate)
- Group 8: Placebo/ Placebo: Participants received matched placebo sterile 0.9% saline IM vaccine at Week 0, 12, 24 and 48.
Period: Main Study (From Week 0 up to Week 96)
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Started | 50 | 49 | 49 | 48 | 49 | 49 | 50 | 49
Completed | 44 | 39 | 44 | 39 | 41 | 43 | 37 | 42
Not Completed | 6 | 10 | 5 | 9 | 8 | 6 | 13 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 5 | 3 | 3 | 2 | 1 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 3 | 4 | 1 | 1 | 2
Not completed — Other | 4 | 2 | 2 | 2 | 1 | 2 | 8 | 2
Period: LTE (After Week 96 up to Week 336)
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Started | 31 | 32 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 29 | 27 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo | Total
Number analyzed (Participants) | 50 | 49 | 49 | 48 | 49 | 49 | 50 | 49 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (7.77) | 29.6 (7.49) | 31.1 (8.22) | 29.6 (7.67) | 30.3 (7.61) | 29.2 (8.73) | 30.3 (7.65) | 29 (8.06) | 29.9 (7.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 28 | 19 | 25 | 19 | 19 | 20 | 181
  Male | 25 | 23 | 21 | 29 | 24 | 30 | 31 | 29 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 2 | 6 | 3 | 5 | 3 | 6 | 35
  Not Hispanic or Latino | 46 | 43 | 46 | 42 | 46 | 44 | 47 | 43 | 357
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 9 | 7 | 9 | 7 | 7 | 8 | 8 | 9 | 64
  Black or African American | 27 | 29 | 27 | 27 | 26 | 26 | 32 | 25 | 219
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 14 | 13 | 11 | 14 | 15 | 13 | 9 | 15 | 104
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  RWANDA | 7 | 7 | 10 | 8 | 9 | 6 | 5 | 6 | 58
  SOUTH AFRICA | 7 | 10 | 5 | 7 | 5 | 7 | 9 | 6 | 56
  THAILAND | 8 | 7 | 7 | 7 | 7 | 7 | 8 | 7 | 58
  UGANDA | 9 | 7 | 8 | 8 | 9 | 10 | 9 | 11 | 71
  UNITED STATES | 19 | 18 | 19 | 18 | 19 | 19 | 19 | 19 | 150

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) Post Vaccination
Description: Solicited local AEs (at injection site) included erythema, induration, swelling, itching and warmth were collected within 7 days after vaccination.
Time Frame: Up to Week 49 (7 days post any dose)
Population: The FAS included all randomized participants with at least one study vaccine administration documented regardless of the occurrence of protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 50 | 49 | 49 | 48 | 49 | 49 | 50 | 49
percentage of participants | 88.0 | 83.7 | 75.5 | 77.1 | 77.6 | 77.6 | 70.0 | 57.1

2. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) Post Vaccination
Description: Solicited systemic AEs included fever (defined as body temperature of 38.0-degree celsius or higher), headache, fatigue, myalgia, nausea, vomiting were collected within 7 days after vaccination.
Time Frame: Up to Week 49 (7 days post any dose)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 50 | 49 | 49 | 48 | 49 | 49 | 50 | 49
percentage of participants | 88.0 | 85.7 | 73.5 | 75.0 | 87.8 | 73.5 | 62.0 | 59.2

3. Primary Outcome: Percentage of Participants With Unsolicited Adverse Events Post Vaccination
Description: Unsolicited AEs were defined as events that participants experienced but were not specifically asked about.
Time Frame: Up to Week 52 (28 days post vaccination)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 50 | 49 | 49 | 48 | 49 | 49 | 50 | 49
percentage of participants | 80.0 | 73.5 | 85.7 | 87.5 | 69.4 | 83.7 | 86.0 | 77.6

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Post Vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. A SAE is any AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Serious adverse events (SAEs) were reported up to Week 336 for Group 1 and 2 and up to Week 96 for the other groups (Group 3, 4, 5, 6, 7, and 8). Other adverse events (AEs) were reported for the main study period up to Week 96 for all the groups
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 50 | 49 | 49 | 48 | 49 | 49 | 50 | 49
Participants | 5 | 2 | 3 | 4 | 4 | 5 | 2 | 5

5. Primary Outcome: Percentage of Responders for Envelop (Env) Clade A, B and C-specific Binding Antibody Titers at Week 28
Description: The Env Clade A (92UG037.1), B (1990a), and C (Con C), (C97ZA.012)- specific binding antibody titer were assessed using enzyme-linked immunosorbent assay (ELISA). The response was defined as post-baseline value greater than (>) lower limit of quantification (LLOQ) if baseline less than (<) LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline greater than or equal to (>=) LLOQ. The lower limits of quantification (LLOQs) for this assay were 625, 156.25, 625, and 156.25 endotoxin units per milliliter (EU/mL) for Clade A (92UG037.1), Clade B (1990a), Clade C (Con C), and Clade C (C97ZA.012) respectively.
Time Frame: Week 28
Population: Per protocol immunogenicity (PPI) analysis set: participants who received at least first 3 vaccines as scheduled, had at least 1 post-vaccination immunogenicity blood draw and not diagnosed with HIV. N(number of participants analyzed): participants who were evaluable for this OM. n(number analyzed): participants evaluable for specified categories.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 49 | 41 | 46 | 44 | 44 | 42 | 44 | 46
percentage of responders
  Clade A (92UG037.1): number analyzed (Participants) | 48 | 41 | 46 | 44 | 43 | 42 | 44 | 46
  Clade A (92UG037.1) | 100.0 [92.6 to 100] | 97.6 [87.14 to 99.94] | 97.8 [88.47 to 99.94] | 95.5 [84.53 to 99.44] | 97.7 [87.71 to 99.94] | 97.6 [87.43 to 99.94] | 95.5 [84.53 to 99.44] | 2.2 [0.06 to 11.53]
  Clade B (1990a): number analyzed (Participants) | 48 | 41 | 46 | 42 | 42 | 42 | 44 | 46
  Clade B (1990a) | 100.0 [92.6 to 100] | 100.0 [91.4 to 100] | 100.0 [92.29 to 100] | 100.0 [91.59 to 100] | 100.0 [91.59 to 100] | 100.0 [91.59 to 100] | 100.0 [91.96 to 100] | 6.5 [1.37 to 17.9]
  Clade C (Con C): number analyzed (Participants) | 47 | 41 | 46 | 44 | 43 | 42 | 44 | 46
  Clade C (Con C) | 100.0 [92.45 to 100] | 100.0 [91.4 to 100] | 100.0 [92.29 to 100] | 95.5 [84.53 to 99.44] | 100.0 [91.78 to 100] | 100.0 [91.59 to 100] | 97.7 [87.98 to 99.94] | 6.5 [1.37 to 17.9]
  Clade C (C97ZA.012): number analyzed (Participants) | 48 | 41 | 46 | 44 | 43 | 42 | 44 | 46
  Clade C (C97ZA.012) | 100 [92.6 to 100] | 100 [91.4 to 100] | 100 [92.29 to 100] | 97.7 [87.98 to 99.94] | 100 [91.59 to 100] | 100 [91.59 to 100] | 100 [91.96 to 100] | 2.2 [0.06 to 11.53]

6. Secondary Outcome: Percentage of Responders for Clade C (C97ZA.012) Env Enzyme-linked Immunosorbent Assay (ELISA) Immunoglobulin G1 (IgG1), IgG2, IgG3 and IgG4 Glycoprotein (gp) 140 Binding Antibody
Description: Vaccine-induced binding antibody IgG1, IgG2, IgG3 and IgG4 subclass responses were investigated using Clade C (C97ZA.012) specific ELISAs. The response was defined as post-baseline value >LLOQ if baseline <LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=LLOQ. The LLOQs for this assay were 12.3, 28.7, 12.4, and 13.2 for IgG1, IgG2, IgG3 and IgG4 respectively. Samples taken after Week 48 (W48) from PPI set, who missed 4th vaccine or deviated schedule were excluded. As planned, the data reported for this endpoint at specified time points only for each reported category.
Time Frame: Week 28, 52 and 96
Population: PPI analysis set. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here 'n' (number analyzed) signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 47 | 41 | 46 | 45 | 42 | 40 | 44 | 45
percentage of responders
  Clade C (C97ZA.012) IgG1 at Week 28 | 78.7 [64.34 to 89.3] | 80.5 [65.13 to 91.18] | 50.0 [34.9 to 65.1] | 82.2 [67.95 to 92] | 61.9 [45.64 to 76.43] | 67.5 [50.87 to 81.43] | 81.8 [67.29 to 91.81] | 0.0 [0.0 to 7.87]
  Clade C (C97ZA.012) IgG1 at Week 52: number analyzed (Participants) | 44 | 38 | 42 | 41 | 39 | 40 | 38 | 40
  Clade C (C97ZA.012) IgG1 at Week 52 | 81.8 [67.29 to 91.81] | 94.7 [82.25 to 99.36] | 59.5 [43.28 to 74.37] | 82.9 [67.94 to 92.85] | 71.8 [55.13 to 85] | 72.5 [56.11 to 85.4] | 89.5 [75.2 to 97.06] | 0 [0 to 8.81]
  Clade C (C97ZA.012) IgG1 at Week 96: number analyzed (Participants) | 41 | 38 | 23 | 21 | 24 | 25 | 24 | 0
  Clade C (C97ZA.012) IgG1 at Week 96 | 36.6 [22.12 to 53.06] | 26.3 [13.4 to 43.1] | 4.3 [0.11 to 21.95] | 38.1 [18.11 to 61.56] | 16.7 [4.74 to 37.38] | 0 [0 to 13.72] | 50.0 [29.12 to 70.88] |
  Clade C (C97ZA.012) IgG2 at Week 28 | 0 [0 to 7.55] | 0 [0 to 8.6] | 2.2 [0.06 to 11.53] | 2.2 [0.06 to 11.77] | 2.4 [0.06 to 12.57] | 0 [0 to 8.81] | 2.3 [0.06 to 12.02] | 0 [0 to 7.87]
  Clade C (C97ZA.012) IgG2 at Week 52: number analyzed (Participants) | 43 | 38 | 42 | 41 | 39 | 40 | 38 | 40
  Clade C (C97ZA.012) IgG2 at Week 52 | 2.3 [0.06 to 12.29] | 0 [0 to 9.25] | 0 [0 to 8.41] | 4.9 [0.6 to 16.53] | 7.7 [1.62 to 20.87] | 0 [0 to 8.81] | 7.9 [1.66 to 21.38] | 0 [0 to 8.81]
  Clade C (C97ZA.012) IgG3 at Week 28: number analyzed (Participants) | 47 | 41 | 46 | 44 | 41 | 39 | 44 | 45
  Clade C (C97ZA.012) IgG3 at Week 28 | 44.7 [30.17 to 59.88] | 29.3 [16.13 to 45.54] | 10.9 [3.62 to 23.57] | 47.7 [32.46 to 63.31] | 29.3 [16.13 to 45.54] | 20.5 [9.3 to 36.46] | 25.0 [13.19 to 40.34] | 0 [0 to 7.87]
  Clade C (C97ZA.012) IgG3 at Week 52: number analyzed (Participants) | 44 | 38 | 42 | 41 | 39 | 39 | 37 | 40
  Clade C (C97ZA.012) IgG3 at Week 52 | 43.2 [28.35 to 58.97] | 42.1 [26.31 to 59.18] | 7.1 [1.5 to 19.48] | 51.2 [35.13 to 67.12] | 35.9 [21.2 to 52.82] | 15.4 [5.86 to 30.53] | 43.2 [27.1 to 60.51] | 0 [0 to 8.81]
  Clade C (C97ZA.012) IgG3 at Week 96: number analyzed (Participants) | 41 | 36 | 25 | 22 | 22 | 24 | 24 | 0
  Clade C (C97ZA.012) IgG3 at Week 96 | 12.2 [4.08 to 26.2] | 8.3 [1.75 to 22.47] | 4.0 [0.1 to 20.35] | 4.5 [0.12 to 22.84] | 13.6 [2.91 to 34.91] | 8.3 [1.03 to 27] | 16.7 [4.74 to 37.38] |
  Clade C (C97ZA.012) IgG4 at Week 28: number analyzed (Participants) | 47 | 41 | 45 | 45 | 42 | 40 | 44 | 45
  Clade C (C97ZA.012) IgG4 at Week 28 | 0 [0 to 7.55] | 0 [0 to 8.6] | 0 [0 to 7.87] | 4.4 [0.54 to 15.15] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 8.04] | 0 [0 to 7.87]
  Clade C (C97ZA.012) IgG4 at Week 52: number analyzed (Participants) | 44 | 38 | 42 | 41 | 39 | 40 | 38 | 40
  Clade C (C97ZA.012) IgG4 at Week 52 | 2.3 [0.06 to 12.02] | 2.6 [0.07 to 13.81] | 0 [0 to 8.41] | 7.3 [1.54 to 19.92] | 0 [0 to 9.03] | 0 [0 to 8.81] | 5.3 [0.64 to 17.75] | 0 [0 to 8.81]

7. Secondary Outcome: Percentage of Responders for Env ELISA Including Consensus C and Mos1 Antigens
Description: The response was defined as post-baseline value >LLOQ if baseline <LLOQ or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=LLOQ. The LLOQ for this assay is a 50 percent (%) inhibitory concentration (IC50) of 20 (fold-dilution). The lower limits of quantification (LLOQs) for this assay were 625 and 78.125 EU/mL for Clade C (Con C) and Mos1 respectively. Samples taken after W48 from PPI set, who missed 4th vaccine or deviated schedule were excluded. As planned, the data reported for this endpoint at specified time points only for each reported category.
Time Frame: Week 28, 52 and 96
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 49 | 41 | 46 | 44 | 44 | 42 | 44 | 46
percentage of responders
  Consensus C (Con C) at Week 28: number analyzed (Participants) | 47 | 41 | 46 | 44 | 43 | 42 | 44 | 46
  Consensus C (Con C) at Week 28 | 100 [92.45 to 100] | 100.0 [91.4 to 100] | 100.0 [92.29 to 100] | 95.5 [84.53 to 99.44] | 100.0 [91.78 to 100] | 100.0 [91.59 to 100] | 97.7 [87.98 to 99.94] | 6.5 [1.37 to 17.9]
  Consensus C (Con C) at Week 52: number analyzed (Participants) | 44 | 40 | 42 | 41 | 40 | 42 | 38 | 42
  Consensus C (Con C) at Week 52 | 100.0 [92.13 to 100] | 100.0 [91.19 to 100] | 100.0 [91.59 to 100] | 95.1 [83.47 to 99.4] | 100.0 [91.19 to 100] | 100.0 [91.59 to 100] | 97.4 [86.19 to 99.93] | 2.4 [0.06 to 12.57]
  Mos1 at Week 28: number analyzed (Participants) | 46 | 40 | 46 | 43 | 43 | 42 | 44 | 46
  Mos1 at Week 28 | 100.0 [92.29 to 100] | 100.0 [91.19 to 100] | 100.0 [92.29 to 100] | 97.7 [87.71 to 99.94] | 100.0 [91.78 to 100] | 100.0 [91.59 to 100] | 97.7 [87.98 to 99.94] | 4.3 [0.53 to 14.84]
  Mos1 at Week 52: number analyzed (Participants) | 44 | 40 | 41 | 40 | 39 | 42 | 36 | 42
  Mos1 at Week 52 | 100.0 [91.96 to 100.0] | 100.0 [91.19 to 100.0] | 100.0 [91.4 to 100.0] | 97.5 [86.84 to 99.94] | 100.0 [90.97 to 100.0] | 100.0 [91.59 to 100.0] | 100.0 [90.26 to 100] | 0 [0 to 8.41]
  Mos1 at Week 96: number analyzed (Participants) | 42 | 38 | 42 | 38 | 39 | 42 | 35 | 40
  Mos1 at Week 96 | 100.0 [91.59 to 100.0] | 100.0 [90.75 to 100.0] | 100.0 [91.59 to 100.0] | 97.4 [86.19 to 99.93] | 100.0 [90.97 to 100.0] | 100.0 [91.59 to 100] | 97.1 [85.08 to 99.93] | 0 [0 to 8.81]

8. Secondary Outcome: Percentage of Responders for Env Antibody-dependent Cellular Phagocytosis (ADCP) gp Antibody
Description: The functionality of vaccine-induced antibody responses was investigated by the determination of ADCP. The response was defined as post-baseline value > limit of detection (LOD) if baseline <LOD or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=LOD. The lower limits of detection (LODs) for this assay were 5.16, 6.43, 6.49, 4.32 and 4.28 (phagocytic score) for Clade A (92UG037.1), Clade B (1990a), Clade C (Con C), Clade C (C97ZA.012), and Mos1, respectively. Samples taken after W48 from PPI set, who missed 4th vaccine or deviated schedule were excluded. As planned, the data reported for this endpoint at specified time points only for each reported category of Clade A, B, C and Mos 1.
Time Frame: Week 16, 26, 28, 52, 78, and 96
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 47 | 41 | 46 | 45 | 42 | 42 | 44 | 46
percentage of responders
  Clade A (92UG037.1) at Week 16: number analyzed (Participants) | 10 | 10 | 10 | 9 | 8 | 6 | 9 | 8
  Clade A (92UG037.1) at Week 16 | 20.0 [2.52 to 55.61] | 20.0 [2.52 to 55.61] | 10.0 [0.25 to 44.5] | 66.7 [29.93 to 92.51] | 0 [0 to 36.94] | 0 [0 to 45.93] | 0 [0 to 33.63] | 0 [0 to 36.94]
  Clade A (92UG037.1) at Week 28 | 36.2 [22.67 to 51.48] | 29.3 [16.13 to 45.54] | 6.5 [1.37 to 17.9] | 46.7 [31.66 to 62.13] | 21.4 [10.3 to 36.81] | 22.5 [10.84 to 38.45] | 9.1 [2.53 to 21.67] | 0 [0 to 7.71]
  Clade B (1990a) at Week 16: number analyzed (Participants) | 10 | 10 | 10 | 9 | 8 | 6 | 9 | 8
  Clade B (1990a) at Week 16 | 50.0 [18.71 to 81.29] | 50.0 [18.71 to 81.29] | 30.0 [6.67 to 65.25] | 66.7 [29.93 to 92.51] | 37.5 [8.52 to 75.51] | 16.7 [0.42 to 64.12] | 33.3 [7.49 to 70.07] | 0 [0 to 36.94]
  Clade B (1990a) at Week 28 | 78.7 [64.34 to 89.3] | 53.7 [37.42 to 69.34] | 37.0 [23.21 to 52.45] | 71.1 [55.69 to 83.63] | 61.9 [45.64 to 76.43] | 72.5 [56.11 to 85.4] | 36.4 [2.41 to 52.23] | 0 [0 to 7.71]
  Clade C (Con C) at Week 16: number analyzed (Participants) | 10 | 10 | 10 | 9 | 8 | 6 | 9 | 8
  Clade C (Con C) at Week 16 | 30.0 [6.67 to 65.25] | 30.0 [6.67 to 65.25] | 0 [0 to 30.85] | 55.6 [21.2 to 86.3] | 37.5 [8.52 to 75.51] | 0 [0 to 45.93] | 11.1 [0.28 to 48.25] | 0 [0 to 36.94]
  Clade C (Con C) at Week 28 | 55.3 [40.12 to 69.83] | 39.0 [24.2 to 55.5] | 41.3 [27 to 56.77] | 53.3 [37.87 to 68.34] | 45.2 [29.85 to 61.33] | 47.5 [31.51 to 63.87] | 43.2 [28.35 to 58.97] | 8.7 [2.42 to 20.79]
  Clade C (C97ZA.012) at Week 16: number analyzed (Participants) | 10 | 10 | 10 | 9 | 8 | 6 | 9 | 8
  Clade C (C97ZA.012) at Week 16 | 20.0 [2.52 to 55.61] | 40.0 [12.16 to 73.76] | 30.0 [6.67 to 65.25] | 44.4 [13.7 to 78.8] | 12.5 [0.32 to 52.65] | 0 [0 to 45.93] | 11.1 [0.28 to 48.25] | 0 [0 to 36.94]
  Clade C (C97ZA.012) at Week 26: number analyzed (Participants) | 46 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (C97ZA.012) at Week 26 | 93.5 [82.1 to 98.63] |  |  |  |  |  |  |
  Clade C (C97ZA.012) at Week 28 | 72.3 [57.36 to 84.38] | 53.7 [37.42 to 69.34] | 19.6 [9.36 to 33.91] | 57.8 [42.15 to 72.34] | 50.0 [34.19 to 65.81] | 37.5 [22.73 to 54.2] | 45.5 [30.39 to 61.15] | 0 [0 to 7.71]
  Clade C (C97ZA.012) at Week 52: number analyzed (Participants) | 45 | 39 | 42 | 41 | 40 | 42 | 38 | 41
  Clade C (C97ZA.012) at Week 52 | 80.0 [65.4 to 90.42] | 64.1 [47.18 to 78.8] | 23.8 [12.05 to 39.45] | 70.7 [54.46 to 83.87] | 60.0 [43.33 to 75.14] | 21.4 [10.3 to 36.81] | 71.1 [54.1 to 84.58] | 0 [0 to 8.6]
  Clade C (C97ZA.012) at Week 78: number analyzed (Participants) | 44 | 39 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (C97ZA.012) at Week 78 | 29.5 [16.76 to 45.2] | 15.4 [5.86 to 30.53] |  |  |  |  |  |
  Clade C (C97ZA.012) at Week 96: number analyzed (Participants) | 42 | 38 | 25 | 22 | 24 | 25 | 24 | 0
  Clade C (C97ZA.012) at Week 96 | 9.5 [2.66 to 22.62] | 10.5 [2.94 to 24.8] | 0 [0 to 13.72] | 18.2 [5.19 to 40.28] | 4.2 [0.11 to 21.12] | 0 [0 to 13.72] | 12.5 [2.66 to 32.36] |
  Mos1 at Week 16: number analyzed (Participants) | 10 | 10 | 10 | 9 | 8 | 6 | 9 | 8
  Mos1 at Week 16 | 90.0 [55.5 to 99.75] | 90.0 [55.5 to 99.75] | 70.0 [34.75 to 93.33] | 77.8 [39.99 to 97.19] | 100.0 [63.06 to 100.0] | 83.3 [35.88 to 99.58] | 88.9 [51.75 to 99.72] | 0 [0 to 36.94]
  Mos1 at Week 28 | 95.7 [85.46 to 99.48] | 87.8 [73.8 to 95.92] | 84.8 [71.13 to 93.66] | 93.3 [81.73 to 98.6] | 92.9 [80.52 to 98.5] | 92.5 [79.61 to 98.43] | 86.4 [72.65 to 94.83] | 0 [0 to 7.71]

9. Secondary Outcome: Percentage of Responders for Human Immunodeficiency Virus Neutralizing Antibody (HIV nAb)
Description: The functionality of vaccine-induced antibody responses was investigated by the determination of nAb activity in a virus neutralization assay (VNA) using TZM-bl cells and Env-pseudotyped viruses. The response was defined as post-baseline value >LLOQ. The LLOQ for this assay is an inhibitory concentration (IC50) of 20 (fold-dilution). Data reported for the responses against Tier 1 HIV strain Clade C (MW965.26) was reported. Samples taken after W48 from PPI set, who missed 4th vaccine or deviated schedule were excluded. As planned, the data reported for this endpoint at specified time points only for each reported category.
Time Frame: Week 28 and 52
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 48 | 41 | 46 | 45 | 44 | 42 | 44 | 46
percentage of responders
  Clade C (MW965.26) Tier 1 at Week 28: number analyzed (Participants) | 48 | 41 | 46 | 45 | 44 | 41 | 44 | 46
  Clade C (MW965.26) Tier 1 at Week 28 | 54.2 [39.17 to 68.63] | 41.5 [26.32 to 57.89] | 21.7 [10.95 to 36.36] | 51.1 [35.77 to 66.3] | 43.2 [28.35 to 58.97] | 36.6 [22.12 to 53.06] | 29.5 [16.76 to 45.2] | 2.2 [0.06 to 11.53]
  Clade C (MW965.26) Tier 1 at Week 52: number analyzed (Participants) | 45 | 38 | 42 | 41 | 40 | 42 | 38 | 41
  Clade C (MW965.26) Tier 1 at Week 52 | 75.6 [60.46 to 87.12] | 65.8 [48.65 to 80.37] | 11.9 [3.98 to 25.63] | 73.2 [57.06 to 85.78] | 52.5 [36.13 to 68.49] | 45.2 [29.85 to 61.33] | 68.4 [51.35 to 82.5] | 2.4 [0.06 to 12.86]

10. Secondary Outcome: Percentage of Responders for Binding Antibody Multiplex Assay (BAMA) IgG1-IgG4 and IgA and IgG-t Breadth Antibody
Description: The human immunodeficiency virus (HIV)-1 BAMA employs flow-cytometric-based technology that also utilizes antibody and antigen interactions to test for the presence of specific antibodies in an unknown sample with the added advantage of multiplexing the antigens of interest. Positive and negative control standards were run with each assay to ensure specificity. The positivity threshold was determined per antigen based on the plus (+) 3 standard deviation (SD) on the non-specific background. Sample values had to be greater than or equal to this value and had to be 3-fold over the baseline values with a minimum median fluorescent intensities (MFI) value of 100. Samples taken after W48 from PPI set, who missed 4th vaccine or deviated schedule were excluded. As planned, the data reported for this endpoint at specified time points only for each reported category.
Time Frame: Week 16, 28, 52, 78, and 96
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 48 | 40 | 46 | 44 | 44 | 44 | 43 | 45
percentage of responders
  HIV ENV Con S gp140 CFI(Clade M)IgG1 Ab Week(W)16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con S gp140 CFI(Clade M)IgG1 Ab Week(W)16 | 76.6 [61.97 to 87.7] |  |  |  |  |  |  |
  HIV ENV Con S gp140 CFI (Clade M) IgG1 Ab at W28: number analyzed (Participants) | 48 | 37 | 46 | 44 | 41 | 41 | 43 | 45
  HIV ENV Con S gp140 CFI (Clade M) IgG1 Ab at W28 | 95.8 [85.75 to 99.49] | 94.6 [81.81 to 99.34] | 76.1 [61.23 to 87.41] | 90.9 [78.33 to 97.47] | 97.6 [87.14 to 99.94] | 95.1 [83.47 to 99.4] | 88.4 [74.92 to 96.11] | 0 [0 to 7.87]
  HIV ENV Con S gp140 CFI (Clade M) IgG1 Ab at W52: number analyzed (Participants) | 45 | 34 | 42 | 40 | 37 | 41 | 36 | 41
  HIV ENV Con S gp140 CFI (Clade M) IgG1 Ab at W52 | 95.6 [84.85 to 99.46] | 97.1 [84.67 to 99.93] | 61.9 [45.64 to 76.43] | 92.5 [79.61 to 98.43] | 100.0 [90.51 to 100.0] | 80.5 [65.13 to 91.18] | 94.4 [81.34 to 99.32] | 0 [0 to 8.6]
  HIV ENV Con 6 gp120/B (Clade M) IgG1 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con 6 gp120/B (Clade M) IgG1 Ab at W16 | 14.9 [6.2 to 28.31] |  |  |  |  |  |  |
  HIV ENV Con 6 gp120/B (Clade M) IgG1 Ab at W28: number analyzed (Participants) | 48 | 37 | 46 | 44 | 41 | 41 | 43 | 45
  HIV ENV Con 6 gp120/B (Clade M) IgG1 Ab at W28 | 60.4 [45.27 to 74.23] | 40.5 [24.75 to 57.9] | 15.2 [6.34 to 28.87] | 59.1 [43.25 to 73.66] | 39.0 [24.2 to 55.5] | 39.0 [24.2 to 55.5] | 23.3 [11.76 to 38.63] | 0 [0 to 7.87]
  HIV ENV Con 6 gp120/B (Clade M) IgG1 Ab at W52: number analyzed (Participants) | 45 | 34 | 42 | 40 | 37 | 41 | 36 | 41
  HIV ENV Con 6 gp120/B (Clade M) IgG1 Ab at W52 | 60.0 [44.33 to 74.3] | 44.1 [27.19 to 62.11] | 11.9 [3.98 to 25.63] | 62.5 [45.8 to 77.27] | 35.1 [20.21 to 52.54] | 19.5 [8.82 to 34.87] | 22.2 [10.12 to 39.15] | 0 [0 to 8.6]
  HIV ENV gp41 IgG1 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp41 IgG1 Ab at W16 | 59.6 [44.27 to 73.63] |  |  |  |  |  |  |
  HIV ENV gp41 IgG1 Ab at W28: number analyzed (Participants) | 48 | 37 | 46 | 44 | 41 | 41 | 43 | 45
  HIV ENV gp41 IgG1 Ab at W28 | 95.8 [85.75 to 99.49] | 94.6 [81.81 to 99.34] | 78.3 [63.64 to 89.05] | 90.9 [78.33 to 97.47] | 97.6 [87.14 to 99.94] | 82.9 [67.94 to 92.85] | 95.3 [84.19 to 99.43] | 0 [0 to 7.87]
  HIV ENV gp41 IgG1 Ab at W52: number analyzed (Participants) | 45 | 34 | 42 | 40 | 37 | 41 | 36 | 41
  HIV ENV gp41 IgG1 Ab at W52 | 95.6 [84.85 to 99.46] | 97.1 [84.67 to 99.93] | 61.9 [45.64 to 76.43] | 92.5 [79.61 to 98.43] | 97.3 [85.84 to 99.93] | 68.3 [51.91 to 81.92] | 97.2 [85.47 to 99.93] | 0 [0 to 8.6]
  HIV ENV 1086C_D7 gp120 (Clade C) IgG1 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_D7 gp120 (Clade C) IgG1 Ab at W16 | 40.4 [26.37 to 55.73] |  |  |  |  |  |  |
  HIV ENV 1086C_D7 gp120 (Clade C) IgG1 Ab at W28: number analyzed (Participants) | 48 | 37 | 46 | 44 | 41 | 41 | 43 | 45
  HIV ENV 1086C_D7 gp120 (Clade C) IgG1 Ab at W28 | 85.4 [72.24 to 93.93] | 70.3 [53.02 to 84.13] | 56.5 [41.11 to 71.07] | 79.5 [64.7 to 90.2] | 87.8 [73.8 to 95.92] | 70.7 [54.46 to 83.87] | 72.1 [56.33 to 84.67] | 0 [0 to 7.87]
  HIV ENV 1086C_D7 gp120 (Clade C) IgG1 Ab at W52: number analyzed (Participants) | 45 | 34 | 42 | 40 | 37 | 41 | 36 | 41
  HIV ENV 1086C_D7 gp120 (Clade C) IgG1 Ab at W52 | 80.0 [65.4 to 90.42] | 79.4 [62.1 to 91.3] | 35.7 [21.55 to 51.97] | 82.5 [67.22 to 92.66] | 83.8 [67.99 to 93.81] | 46.3 [30.66 to 62.58] | 83.3 [67.19 to 93.63] | 0 [0 to 8.6]
  HIV ENV 1086C gp140 (Clade C) IgG1 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C gp140 (Clade C) IgG1 Ab at W16 | 74.5 [59.65 to 86.06] |  |  |  |  |  |  |
  HIV ENV 1086C gp140 (Clade C) IgG1 Ab at W28: number analyzed (Participants) | 48 | 37 | 46 | 44 | 41 | 41 | 43 | 45
  HIV ENV 1086C gp140 (Clade C) IgG1 Ab at W28 | 93.8 [82.8 to 98.69] | 94.6 [81.81 to 99.34] | 76.1 [61.23 to 87.41] | 90.9 [78.33 to 97.47] | 100.0 [91.4 to 100.0] | 100.0 [91.4 to 100.0] | 86.0 [72.07 to 94.7] | 0 [0 to 7.87]
  HIV ENV 1086C gp140 (Clade C) IgG1 Ab at W52: number analyzed (Participants) | 45 | 34 | 42 | 40 | 37 | 41 | 36 | 41
  HIV ENV 1086C gp140 (Clade C) IgG1 Ab at W52 | 95.6 [84.85 to 99.46] | 97.1 [84.67 to 99.93] | 76.2 [60.55 to 87.95] | 92.5 [79.61 to 98.43] | 97.3 [85.84 to 99.93] | 90.2 [76.87 to 97.28] | 94.4 [81.34 to 99.32] | 0 [0 to 8.6]
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG1 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG1 Ab at W16 | 6.4 [1.34 to 17.54] |  |  |  |  |  |  |
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG1 Ab at W28: number analyzed (Participants) | 48 | 37 | 46 | 44 | 41 | 41 | 43 | 45
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG1 Ab at W28 | 16.7 [7.48 to 30.22] | 10.8 [3.03 to 25.42] | 2.2 [0.06 to 11.53] | 18.2 [8.19 to 32.71] | 19.5 [8.82 to 34.87] | 4.9 [0.6 to 16.53] | 7.0 [1.46 to 19.06] | 0 [0 to 7.87]
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG1 Ab at W52: number analyzed (Participants) | 45 | 34 | 42 | 40 | 37 | 41 | 36 | 41
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG1 Ab at W52 | 20.0 [9.58 to 34.6] | 8.8 [1.86 to 23.68] | 4.8 [0.58 to 16.16] | 25.0 [12.69 to 41.2] | 13.5 [4.54 to 28.77] | 9.8 [2.72 to 23.13] | 13.9 [4.67 to 29.5] | 0 [0 to 8.6]
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG1 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG1 Ab at W16 | 14.9 [6.2 to 28.31] |  |  |  |  |  |  |
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG1 Ab at W28: number analyzed (Participants) | 48 | 37 | 46 | 44 | 41 | 41 | 43 | 45
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG1 Ab at W28 | 29.2 [16.95 to 44.06] | 27.0 [13.79 to 44.12] | 10.9 [3.62 to 23.57] | 20.5 [9.8 to 35.3] | 22.0 [10.56 to 37.61] | 7.3 [1.54 to 19.92] | 7.0 [1.46 to 19.06] | 0 [0 to 7.87]
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG1 Ab at W52: number analyzed (Participants) | 45 | 34 | 42 | 40 | 37 | 41 | 36 | 41
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG1 Ab at W52 | 13.3 [5.05 to 26.79] | 14.7 [4.95 to 31.06] | 9.5 [2.66 to 22.62] | 22.5 [10.84 to 38.45] | 13.5 [4.54 to 28.77] | 0 [0 to 8.6] | 13.9 [4.67 to 29.5] | 2.4 [0.06 to 12.86]
  HIV ENV Con S gp140 CFI (Clade M) IgG2 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con S gp140 CFI (Clade M) IgG2 Ab at W16 | 0 [0 to 7.4] |  |  |  |  |  |  |
  HIV ENV Con S gp140 CFI (Clade M) IgG2 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 42 | 40 | 43 | 45
  HIV ENV Con S gp140 CFI (Clade M) IgG2 Ab at W28 | 2.1 [0.05 to 11.07] | 0 [0 to 8.81] | 0 [0 to 7.71] | 0 [0 to 8.22] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 8.22] | 0 [0 to 7.87]
  HIV ENV Con S gp140 CFI (Clade M) IgG2 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 40 | 37 | 41 | 37 | 41
  HIV ENV Con S gp140 CFI (Clade M) IgG2 Ab at W52 | 2.2 [0.06 to 11.77] | 0 [0 to 9.49] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 9.49] | 0 [0 to 8.6] | 0 [0 to 9.49] | 0 [0 to 8.6]
  HIV ENV Con 6 gp120/B (Clade M) IgG2 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con 6 gp120/B (Clade M) IgG2 Ab at W16 | 0 [0 to 7.4] |  |  |  |  |  |  |
  HIV ENV Con 6 gp120/B (Clade M) IgG2 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 42 | 40 | 43 | 45
  HIV ENV Con 6 gp120/B (Clade M) IgG2 Ab at W28 | 0 [0 to 7.4] | 0 [0 to 8.81] | 0 [0 to 7.71] | 0 [0 to 8.22] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 8.22] | 0 [0 to 7.87]
  HIV ENV Con 6 gp120/B (Clade M) IgG2 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 40 | 37 | 41 | 37 | 41
  HIV ENV Con 6 gp120/B (Clade M) IgG2 Ab at W52 | 0 [0 to 7.87] | 0 [0 to 9.49] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 9.49] | 0 [0 to 8.6] | 0 [0 to 9.49] | 0 [0 to 8.6]
  HIV ENV gp41 IgG2 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp41 IgG2 Ab at W16 | 0 [0 to 7.4] |  |  |  |  |  |  |
  HIV ENV gp41 IgG2 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 42 | 40 | 43 | 45
  HIV ENV gp41 IgG2 Ab at W28 | 2.1 [0.05 to 11.07] | 0 [0 to 8.81] | 0 [0 to 7.71] | 2.3 [0.06 to 12.29] | 2.4 [0.06 to 12.57] | 0 [0 to 8.81] | 0 [0 to 8.22] | 0 [0 to 7.87]
  HIV ENV gp41 IgG2 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 40 | 37 | 41 | 37 | 41
  HIV ENV gp41 IgG2 Ab at W52 | 0 [0 to 7.87] | 2.7 [0.07 to 14.16] | 0 [0 to 8.41] | 5.0 [0.61 to 16.92] | 0 [0 to 9.49] | 0 [0 to 8.6] | 0 [0 to 9.49] | 0 [0 to 8.6]
  HIV ENV 1086C_D7 gp120 (Clade C) IgG2 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_D7 gp120 (Clade C) IgG2 Ab at W16 | 2.1 [0.05 to 11.07] |  |  |  |  |  |  |
  HIV ENV 1086C_D7 gp120 (Clade C) IgG2 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 42 | 40 | 43 | 45
  HIV ENV 1086C_D7 gp120 (Clade C) IgG2 Ab at W28 | 2.1 [0.05 to 11.07] | 0 [0 to 8.81] | 0 [0 to 7.71] | 2.3 [0.06 to 12.29] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 8.22] | 0 [0 to 7.87]
  HIV ENV 1086C_D7 gp120 (Clade C) IgG2 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 40 | 37 | 41 | 37 | 41
  HIV ENV 1086C_D7 gp120 (Clade C) IgG2 Ab at W52 | 0 [0 to 7.87] | 0 [0 to 9.49] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 9.49] | 0 [0 to 8.6] | 0 [0 to 9.49] | 0 [0 to 8.6]
  HIV ENV 1086C gp140 (Clade C) IgG2 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C gp140 (Clade C) IgG2 Ab at W16 | 2.1 [0.05 to 11.07] |  |  |  |  |  |  |
  HIV ENV 1086C gp140 (Clade C) IgG2 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 42 | 40 | 41 | 45
  HIV ENV 1086C gp140 (Clade C) IgG2 Ab at W28 | 2.1 [0.05 to 11.07] | 0 [0 to 8.81] | 0 [0 to 7.71] | 2.3 [0.06 to 12.29] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 8.22] | 0 [0 to 7.87]
  HIV ENV 1086C gp140 (Clade C) IgG2 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 40 | 37 | 41 | 37 | 41
  HIV ENV 1086C gp140 (Clade C) IgG2 Ab at W52 | 2.2 [0.06 to 11.77] | 0 [0 to 9.49] | 0 [0 to 8.41] | 2.5 [0.06 to 13.16] | 2.7 [0.07 to 14.16] | 0 [0 to 8.6] | 0 [0 to 9.49] | 0 [0 to 8.6]
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG2 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG2 Ab at W16 | 0 [0 to 7.4] |  |  |  |  |  |  |
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG2 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 42 | 40 | 43 | 45
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG2 Ab at W28 | 0 [0 to 7.4] | 0 [0 to 8.81] | 0 [0 to 7.71] | 0 [0 to 8.22] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 8.22] | 0 [0 to 7.87]
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG2 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 40 | 37 | 41 | 37 | 41
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG2 Ab at W52 | 0 [0 to 7.87] | 0 [0 to 9.49] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 9.49] | 0 [0 to 8.6] | 0 [0 to 9.49] | 0 [0 to 8.6]
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG2 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG2 Ab at W16 | 0 [0 to 7.4] |  |  |  |  |  |  |
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG2 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 42 | 40 | 43 | 45
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG2 Ab at W28 | 0 [0 to 7.4] | 2.5 [0.06 to 13.16] | 0 [0 to 7.71] | 0 [0 to 8.22] | 2.4 [0.06 to 12.57] | 0 [0 to 8.81] | 0 [0 to 8.22] | 0 [0 to 7.87]
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG2 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 40 | 37 | 41 | 37 | 41
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG2 Ab at W52 | 0 [0 to 7.87] | 0 [0 to 9.49] | 0 [0 to 8.41] | 0 [0 to 8.81] | 0 [0 to 9.49] | 0 [0 to 8.6] | 0 [0 to 9.49] | 0 [0 to 8.6]
  HIV ENV Con S gp140 CFI (Clade M) IgG3 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con S gp140 CFI (Clade M) IgG3 Ab at W16 | 61.7 [46.38 to 75.49] |  |  |  |  |  |  |
  HIV ENV Con S gp140 CFI (Clade M) IgG3 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 43 | 41 | 43 | 45
  HIV ENV Con S gp140 CFI (Clade M) IgG3 Ab at W28 | 75.0 [60.4 to 86.36] | 47.5 [31.51 to 63.87] | 34.8 [21.35 to 50.25] | 76.7 [61.37 to 88.24] | 79.1 [63.96 to 89.96] | 58.5 [42.11 to 73.68] | 67.4 [51.46 to 80.92] | 0 [0 to 7.87]
  HIV ENV Con S gp140 CFI (Clade M) IgG3 Ab at W52: number analyzed (Participants) | 43 | 37 | 41 | 38 | 39 | 41 | 37 | 39
  HIV ENV Con S gp140 CFI (Clade M) IgG3 Ab at W52 | 76.7 [61.37 to 88.24] | 59.5 [42.1 to 75.25] | 56.1 [39.75 to 71.53] | 78.9 [62.68 to 90.45] | 82.1 [66.47 to 92.46] | 48.8 [32.88 to 64.87] | 81.1 [64.84 to 92.04] | 7.7 [1.62 to 20.87]
  HIV ENV Con S gp140 CFI (Clade M) IgG3 Ab at W78: number analyzed (Participants) | 43 | 38 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con S gp140 CFI (Clade M) IgG3 Ab at W78 | 53.5 [37.65 to 68.82] | 28.9 [15.42 to 45.9] |  |  |  |  |  |
  HIV ENV Con S gp140 CFI (Clade M) IgG3 Ab at W96: number analyzed (Participants) | 41 | 35 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con S gp140 CFI (Clade M) IgG3 Ab at W96 | 48.8 [32.88 to 64.87] | 34.3 [19.13 to 52.21] |  |  |  |  |  |
  HIV ENV Con 6 gp120/B (Clade M) IgG3 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con 6 gp120/B (Clade M) IgG3 Ab at W16 | 31.9 [19.09 to 47.12] |  |  |  |  |  |  |
  HIV ENV Con 6 gp120/B (Clade M) IgG3 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 43 | 41 | 43 | 45
  HIV ENV Con 6 gp120/B (Clade M) IgG3 Ab at W28 | 31.3 [18.66 to 46.25] | 22.5 [10.84 to 38.45] | 10.9 [3.62 to 23.57] | 32.6 [19.08 to 48.54] | 23.3 [11.76 to 38.63] | 22.0 [10.56 to 37.61] | 11.6 [3.89 to 25.08] | 0 [0 to 7.87]
  HIV ENV Con 6 gp120/B (Clade M) IgG3 Ab at W52: number analyzed (Participants) | 43 | 37 | 41 | 38 | 39 | 41 | 37 | 39
  HIV ENV Con 6 gp120/B (Clade M) IgG3 Ab at W52 | 48.8 [33.31 to 64.54] | 27.0 [13.79 to 44.12] | 17.1 [7.15 to 32.06] | 47.4 [30.98 to 64.18] | 46.2 [30.09 to 62.82] | 31.7 [18.08 to 48.09] | 24.3 [11.77 to 41.2] | 2.6 [0.06 to 13.48]
  HIV ENV Con 6 gp120/B (Clade M) IgG3 Ab at W78: number analyzed (Participants) | 43 | 38 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con 6 gp120/B (Clade M) IgG3 Ab at W78 | 14.0 [5.3 to 27.93] | 7.9 [1.66 to 21.38] |  |  |  |  |  |
  HIV ENV Con 6 gp120/B (Clade M) IgG3 Ab at W96: number analyzed (Participants) | 41 | 35 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con 6 gp120/B (Clade M) IgG3 Ab at W96 | 17.1 [7.15 to 32.06] | 8.6 [1.8 to 23.06] |  |  |  |  |  |
  HIV ENV gp41 IgG3 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp41 IgG3 Ab at W16 | 25.5 [13.94 to 40.35] |  |  |  |  |  |  |
  HIV ENV gp41 IgG3 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 43 | 41 | 43 | 45
  HIV ENV gp41 IgG3 Ab at W28 | 52.1 [37.19 to 66.71] | 45.0 [29.26 to 61.51] | 13.0 [4.94 to 26.26] | 55.8 [39.88 to 70.92] | 58.1 [42.13 to 72.99] | 26.8 [14.22 to 42.94] | 46.5 [31.18 to 62.35] | 0 [0 to 7.87]
  43HIV ENV gp41 IgG3 Ab at W52: number analyzed (Participants) | 43 | 37 | 41 | 38 | 39 | 41 | 41 | 39
  43HIV ENV gp41 IgG3 Ab at W52 | 67.4 [51.46 to 80.92] | 54.1 [36.92 to 70.51] | 14.6 [5.57 to 29.17] | 73.7 [56.9 to 86.6] | 79.5 [63.54 to 90.7] | 26.8 [14.22 to 42.94] | 67.6 [50.21 to 81.99] | 7.7 [1.62 to 20.87]
  HIV ENV gp41 IgG3 Ab at W78: number analyzed (Participants) | 43 | 38 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp41 IgG3 Ab at W78 | 34.9 [21.01 to 50.93] | 23.7 [11.44 to 40.24] |  |  |  |  |  |
  HIV ENV gp41 IgG3 Ab at W96: number analyzed (Participants) | 41 | 35 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp41 IgG3 Ab at W96 | 31.7 [18.08 to 48.09] | 22.9 [10.42 to 40.14] |  |  |  |  |  |
  HIV ENV 1086C_D7 gp120 (Clade C) IgG3 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_D7 gp120 (Clade C) IgG3 Ab at W16 | 68.1 [52.88 to 80.91] |  |  |  |  |  |  |
  HIV ENV 1086C_D7 gp120 (Clade C) IgG3 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 43 | 41 | 43 | 45
  HIV ENV 1086C_D7 gp120 (Clade C) IgG3 Ab at W28 | 66.7 [51.59 to 79.6] | 50.0 [33.8 to 66.2] | 39.1 [25.09 to 54.63] | 65.1 [49.07 to 78.99] | 65.1 [49.07 to 78.99] | 58.5 [42.11 to 73.68] | 53.5 [37.65 to 68.82] | 0 [0 to 7.87]
  HIV ENV 1086C_D7 gp120 (Clade C) IgG3 Ab at W52: number analyzed (Participants) | 43 | 37 | 41 | 38 | 39 | 41 | 37 | 39
  HIV ENV 1086C_D7 gp120 (Clade C) IgG3 Ab at W52 | 76.7 [61.37 to 88.24] | 67.6 [50.21 to 81.99] | 51.2 [35.13 to 67.12] | 78.9 [62.68 to 90.45] | 82.1 [66.47 to 92.46] | 58.5 [42.11 to 73.68] | 75.7 [58.8 to 88.23] | 2.6 [0.06 to 13.48]
  HIV ENV 1086C_D7 gp120 (Clade C) IgG3 Ab at W78: number analyzed (Participants) | 43 | 38 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_D7 gp120 (Clade C) IgG3 Ab at W78 | 53.5 [37.65 to 68.82] | 39.5 [24.04 to 56.61] |  |  |  |  |  |
  HIV ENV 1086C_D7 gp120 (Clade C) IgG3 Ab at W96: number analyzed (Participants) | 41 | 35 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_D7 gp120 (Clade C) IgG3 Ab at W96 | 48.8 [32.88 to 64.87] | 37.1 [21.47 to 55.08] |  |  |  |  |  |
  HIV ENV 1086C gp140 (Clade C) IgG3 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C gp140 (Clade C) IgG3 Ab at W16 | 74.5 [59.65 to 86.06] |  |  |  |  |  |  |
  HIV ENV 1086C gp140 (Clade C) IgG3 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 43 | 41 | 43 | 45
  HIV ENV 1086C gp140 (Clade C) IgG3 Ab at W28 | 83.3 [69.78 to 92.52] | 60.0 [43.33 to 75.14] | 67.4 [51.98 to 80.47] | 86.0 [72.07 to 94.7] | 86.0 [72.07 to 94.7] | 75.6 [59.7 to 87.64] | 76.7 [61.37 to 88.24] | 0 [0 to 7.87]
  HIV ENV 1086C gp140 (Clade C) IgG3 Ab at W52: number analyzed (Participants) | 43 | 37 | 41 | 38 | 39 | 41 | 37 | 39
  HIV ENV 1086C gp140 (Clade C) IgG3 Ab at W52 | 81.4 [66.6 to 91.61] | 70.3 [53.02 to 84.13] | 65.9 [49.41 to 79.92] | 86.8 [71.91 to 95.59] | 87.2 [72.57 to 95.7] | 61.0 [44.5 to 75.8] | 83.8 [67.99 to 93.81] | 2.6 [0.06 to 13.48]
  HIV ENV 1086C gp140 (Clade C) IgG3 Ab at W78: number analyzed (Participants) | 43 | 38 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C gp140 (Clade C) IgG3 Ab at W78 | 55.8 [39.88 to 70.92] | 36.8 [21.81 to 54.01] |  |  |  |  |  |
  HIV ENV 1086C gp140 (Clade C) IgG3 Ab at W96: number analyzed (Participants) | 41 | 35 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C gp140 (Clade C) IgG3 Ab at W96 | 46.3 [30.66 to 62.58] | 31.4 [16.85 to 49.29] |  |  |  |  |  |
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG3 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG3 Ab at W16 | 12.8 [4.83 to 25.74] |  |  |  |  |  |  |
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG3 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 43 | 41 | 43 | 45
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG3 Ab at W28 | 18.8 [8.95 to 32.63] | 12.5 [4.19 to 26.8] | 6.5 [1.37 to 17.9] | 23.3 [11.76 to 38.63] | 16.3 [6.81 to 30.7] | 14.6 [5.57 to 29.17] | 16.3 [6.81 to 30.7] | 0 [0 to 7.87]
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG3 Ab at W52: number analyzed (Participants) | 43 | 37 | 41 | 38 | 39 | 41 | 37 | 39
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG3 Ab at W52 | 25.6 [13.52 to 41.17] | 10.8 [3.03 to 25.42] | 9.8 [2.72 to 23.13] | 28.9 [15.42 to 45.9] | 15.4 [5.86 to 30.53] | 9.8 [2.72 to 23.13] | 16.2 [6.19 to 32.01] | 2.6 [0.06 to 13.48]
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG3 Ab at W78: number analyzed (Participants) | 43 | 38 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG3 Ab at W78 | 4.7 [0.57 to 15.81] | 2.6 [0.07 to 13.81] |  |  |  |  |  |
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG3 Ab at W96: number analyzed (Participants) | 41 | 35 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG3 Ab at W96 | 9.8 [2.72 to 23.13] | 8.6 [1.8 to 23.06] |  |  |  |  |  |
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG3 Ab at W16: number analyzed (Participants) | 47 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG3 Ab at W16 | 14.9 [6.2 to 28.31] |  |  |  |  |  |  |
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG3 Ab at W28: number analyzed (Participants) | 48 | 40 | 45 | 43 | 43 | 41 | 43 | 45
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG3 Ab at W28 | 12.5 [4.73 to 25.25] | 12.5 [4.19 to 26.8] | 11.1 [3.71 to 24.05] | 18.6 [8.39 to 33.4] | 11.6 [3.89 to 25.08] | 12.2 [4.08 to 26.2] | 7.0 [1.46 to 19.06] | 0 [0 to 7.87]
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG3 Ab at W52: number analyzed (Participants) | 43 | 37 | 40 | 38 | 39 | 40 | 37 | 39
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG3 Ab at W52 | 18.6 [8.39 to 33.4] | 10.8 [3.03 to 25.42] | 5.0 [0.61 to 16.92] | 28.9 [15.42 to 45.9] | 7.7 [1.62 to 20.87] | 7.5 [1.57 to 20.39] | 10.8 [3.03 to 25.42] | 2.6 [0.06 to 13.48]
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG3 Ab at W78: number analyzed (Participants) | 43 | 38 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG3 Ab at W78 | 2.3 [0.06 to 12.29] | 2.6 [0.07 to 13.81] |  |  |  |  |  |
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG3 Ab at W96: number analyzed (Participants) | 41 | 35 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG3 Ab at W96 | 2.4 [0.06 to 12.86] | 2.9 [0.07 to 14.92] |  |  |  |  |  |
  HIV ENV Con S gp140 CFI (Clade M) IgG4 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con S gp140 CFI (Clade M) IgG4 Ab at W16 | 10.4 [3.47 to 22.66] |  |  |  |  |  |  |
  HIV ENV Con S gp140 CFI (Clade M) IgG4 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 44 | 41 | 43 | 45
  HIV ENV Con S gp140 CFI (Clade M) IgG4 Ab at W28 | 12.5 [4.73 to 25.25] | 10.0 [2.79 to 23.66] | 13.0 [4.94 to 26.26] | 9.3 [2.59 to 22.14] | 9.1 [2.53 to 21.67] | 7.3 [1.54 to 19.92] | 16.3 [6.81 to 30.7] | 0 [0 to 7.87]
  HIV ENV Con S gp140 CFI (Clade M) IgG4 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 38 | 40 | 41 | 37 | 41
  HIV ENV Con S gp140 CFI (Clade M) IgG4 Ab at W52 | 40.0 [25.7 to 55.67] | 29.7 [15.87 to 46.98] | 19.0 [8.6 to 34.12] | 28.9 [15.42 to 45.9] | 20.0 [9.05 to 35.65] | 12.2 [4.08 to 26.2] | 35.1 [20.21 to 52.54] | 0 [0 to 8.6]
  HIV ENV Con 6 gp120/B (Clade M) IgG4 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con 6 gp120/B (Clade M) IgG4 Ab at W16 | 0 [0 to 7.4] |  |  |  |  |  |  |
  HIV ENV Con 6 gp120/B (Clade M) IgG4 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 44 | 41 | 43 | 45
  HIV ENV Con 6 gp120/B (Clade M) IgG4 Ab at W28 | 2.1 [0.05 to 11.07] | 2.5 [0.06 to 13.16] | 0 [0 to 7.71] | 4.7 [0.57 to 15.81] | 0 [0 to 8.04] | 0 [0 to 8.6] | 7.0 [1.46 to 19.06] | 0 [0 to 7.87]
  HIV ENV Con 6 gp120/B (Clade M) IgG4 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 38 | 40 | 41 | 37 | 41
  HIV ENV Con 6 gp120/B (Clade M) IgG4 Ab at W52 | 15.6 [6.49 to 29.46] | 10.8 [3.03 to 25.42] | 2.4 [0.06 to 12.57] | 18.4 [7.74 to 34.33] | 5.0 [0.61 to 16.92] | 0 [0 to 8.6] | 8.1 [1.7 to 21.91] | 0 [0 to 8.6]
  HIV ENV gp41 IgG4 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp41 IgG4 Ab at W16 | 10.4 [3.47 to 22.66] |  |  |  |  |  |  |
  HIV ENV gp41 IgG4 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 44 | 41 | 43 | 45
  HIV ENV gp41 IgG4 Ab at W28 | 33.3 [20.4 to 48.41] | 15.0 [5.71 to 29.84] | 13.0 [4.94 to 26.26] | 25.6 [13.52 to 41.17] | 20.5 [9.8 to 35.3] | 7.3 [1.54 to 19.92] | 34.9 [21.01 to 50.93] | 2.2 [0.06 to 11.77]
  HIV ENV gp41 IgG4 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 38 | 40 | 41 | 37 | 41
  HIV ENV gp41 IgG4 Ab at W52 | 66.7 [51.05 to 80] | 56.8 [39.49 to 72.9] | 16.7 [6.97 to 31.36] | 52.6 [35.82 to 69.02] | 45.0 [29.26 to 61.51] | 7.3 [1.54 to 19.92] | 62.2 [44.76 to 77.54] | 7.3 [1.54 to 19.92]
  HIV ENV 1086C_D7 gp120 (Clade C) IgG4 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_D7 gp120 (Clade C) IgG4 Ab at W16 | 10.4 [3.47 to 22.66] |  |  |  |  |  |  |
  HIV ENV 1086C_D7 gp120 (Clade C) IgG4 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 44 | 44 | 43 | 45
  HIV ENV 1086C_D7 gp120 (Clade C) IgG4 Ab at W28 | 14.6 [6.07 to 27.76] | 7.5 [1.57 to 20.39] | 6.5 [1.37 to 17.9] | 9.3 [2.59 to 22.14] | 6.8 [1.43 to 18.66] | 9.8 [2.72 to 23.13] | 14.0 [5.3 to 27.93] | 0 [0 to 7.87]
  HIV ENV 1086C_D7 gp120 (Clade C) IgG4 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 38 | 40 | 41 | 37 | 41
  HIV ENV 1086C_D7 gp120 (Clade C) IgG4 Ab at W52 | 31.1 [18.17 to 46.65] | 21.6 [9.83 to 38.21] | 9.5 [2.66 to 22.62] | 28.9 [15.42 to 45.9] | 20.0 [9.05 to 35.65] | 12.2 [4.08 to 26.2] | 27.0 [13.79 to 44.12] | 0 [0 to 8.6]
  HIV ENV 1086C gp140 (Clade C) IgG4 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C gp140 (Clade C) IgG4 Ab at W16 | 12.5 [4.73 to 25.25] |  |  |  |  |  |  |
  HIV ENV 1086C gp140 (Clade C) IgG4 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 44 | 41 | 43 | 45
  HIV ENV 1086C gp140 (Clade C) IgG4 Ab at W28 | 18.8 [8.95 to 32.63] | 12.5 [4.19 to 26.8] | 10.9 [3.62 to 23.57] | 9.3 [2.59 to 22.14] | 13.6 [5.17 to 27.35] | 9.8 [2.72 to 23.13] | 16.3 [6.81 to 30.7] | 0 [0 to 7.87]
  HIV ENV 1086C gp140 (Clade C) IgG4 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 38 | 40 | 41 | 37 | 41
  HIV ENV 1086C gp140 (Clade C) IgG4 Ab at W52 | 46.7 [31.66 to 62.13] | 35.1 [20.21 to 52.54] | 16.7 [6.97 to 31.36] | 28.9 [15.42 to 45.9] | 40.0 [24.86 to 56.67] | 22.0 [10.56 to 37.61] | 37.8 [22.46 to 55.24] | 0 [0 to 8.6]
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG4 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG4 Ab at W16 | 0 [0 to 7.4] |  |  |  |  |  |  |
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG4 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 44 | 41 | 43 | 45
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG4 Ab at W28 | 2.1 [0.05 to 11.07] | 2.5 [0.06 to 13.16] | 0 [0 to 7.71] | 4.7 [0.57 to 15.81] | 2.3 [0.06 to 12.02] | 2.4 [0.06 to 12.86] | 2.3 [0.06 to 12.29] | 0 [0 to 7.87]
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG4 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 38 | 40 | 41 | 37 | 41
  HIV ENV 1086C_V1V2 gp70 (Clade C) IgG4 Ab at W52 | 2.2 [0.06 to 11.77] | 5.4 [0.66 to 18.19] | 4.8 [0.58 to 16.16] | 2.6 [0.07 to 13.81] | 2.5 [0.06 to 13.16] | 2.4 [0.06 to 12.86] | 5.4 [0.66 to 18.19] | 0 [0 to 8.6]
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG4 Ab at W16: number analyzed (Participants) | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG4 Ab at W16 | 0 [0 to 7.4] |  |  |  |  |  |  |
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG4 Ab at W28: number analyzed (Participants) | 48 | 40 | 46 | 43 | 44 | 41 | 43 | 45
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG4 Ab at W28 | 0 [0 to 7.4] | 0 [0 to 8.81] | 0 [0 to 7.71] | 2.3 [0.06 to 12.29] | 0 [0 to 8.04] | 0 [0 to 8.6] | 0 [0 to 8.22] | 0 [0 to 7.87]
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG4 Ab at W52: number analyzed (Participants) | 45 | 37 | 42 | 38 | 40 | 41 | 37 | 41
  HIV ENV gp70_B.CaseA_V1V2 (Clade B) IgG4 Ab at W52 | 0 [0 to 7.87] | 2.7 [0.07 to 14.16] | 0 [0 to 8.41] | 5.3 [0.64 to 17.75] | 2.5 [0.06 to 13.16] | 2.4 [0.06 to 12.86] | 2.7 [0.07 to 14.16] | 0 [0 to 8.6]
  HIV ENV Con S gp140 CFI (Clade M) IgA Ab at W16: number analyzed (Participants) | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con S gp140 CFI (Clade M) IgA Ab at W16 | 60.0 [43.33 to 75.14] |  |  |  |  |  |  |
  HIV ENV Con S gp140 CFI (Clade M) IgA Ab at W28: number analyzed (Participants) | 39 | 31 | 36 | 35 | 34 | 38 | 37 | 38
  HIV ENV Con S gp140 CFI (Clade M) IgA Ab at W28 | 76.9 [60.67 to 88.87] | 87.1 [70.17 to 96.37] | 77.8 [60.85 to 89.88] | 82.9 [66.35 to 93.44] | 85.3 [68.94 to 95.05] | 78.9 [62.68 to 90.45] | 83.8 [67.99 to 93.81] | 0 [0 to 9.25]
  HIV ENV Con S gp140 CFI (Clade M) IgA Ab at W52: number analyzed (Participants) | 35 | 25 | 31 | 26 | 26 | 32 | 29 | 32
  HIV ENV Con S gp140 CFI (Clade M) IgA Ab at W52 | 77.1 [59.86 to 89.58] | 92.0 [73.97 to 99.02] | 61.3 [42.19 to 78.15] | 84.6 [65.13 to 95.64] | 69.2 [48.21 to 85.67] | 68.8 [49.99 to 83.88] | 86.2 [68.34 to 96.11] | 0 [0 to 10.89]
  HIV ENV Con 6 gp120/B (Clade M) IgA Ab at W16: number analyzed (Participants) | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV Con 6 gp120/B (Clade M) IgA Ab at W16 | 52.5 [36.13 to 68.49] |  |  |  |  |  |  |
  HIV ENV Con 6 gp120/B (Clade M) IgA Ab at W28: number analyzed (Participants) | 39 | 31 | 36 | 35 | 34 | 38 | 37 | 38
  HIV ENV Con 6 gp120/B (Clade M) IgA Ab at W28 | 59.0 [42.1 to 74.43] | 45.2 [27.32 to 63.97] | 44.4 [27.94 to 61.9] | 45.7 [28.83 to 63.35] | 47.1 [29.78 to 64.87] | 39.5 [24.04 to 56.61] | 48.6 [31.92 to 65.6] | 0 [0 to 9.25]
  HIV ENV Con 6 gp120/B (Clade M) IgA Ab at W52: number analyzed (Participants) | 35 | 25 | 31 | 26 | 26 | 32 | 29 | 32
  HIV ENV Con 6 gp120/B (Clade M) IgA Ab at W52 | 60.0 [42.11 to 76.13] | 40.0 [21.13 to 61.33] | 45.2 [27.32 to 63.97] | 50.0 [29.93 to 70.07] | 42.3 [23.35 to 63.08] | 43.8 [26.36 to 62.34] | 55.2 [35.69 to 73.55] | 0 [0 to 10.89]
  HIV ENV 1086C_D7 gp120 (Clade C) IgA Ab at W16: number analyzed (Participants) | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 1086C_D7 gp120 (Clade C) IgA Ab at W16 | 67.5 [50.87 to 81.43] |  |  |  |  |  |  |
  HIV ENV 1086C_D7 gp120 (Clade C) IgA Ab at W28: number analyzed (Participants) | 39 | 31 | 36 | 35 | 34 | 38 | 37 | 38
  HIV ENV 1086C_D7 gp120 (Clade C) IgA Ab at W28 | 71.8 [55.13 to 85] | 77.4 [58.9 to 90.41] | 61.1 [43.46 to 76.86] | 74.3 [56.74 to 87.51] | 79.4 [62.1 to 91.3] | 68.4 [51.35 to 82.5] | 78.4 [61.79 to 90.17] | 0 [0 to 9.25]
  HIV ENV 1086C_D7 gp120 (Clade C) IgA Ab at W52: number analyzed (Participants) | 35 | 25 | 31 | 26 | 26 | 32 | 29 | 31
  HIV ENV 1086C_D7 gp120 (Clade C) IgA Ab at W52 | 74.3 [56.74 to 87.51] | 68.0 [46.5 to 85.05] | 41.9 [24.55 to 60.92] | 76.9 [56.35 to 91.03] | 73.1 [52.21 to 88.43] | 59.4 [40.64 to 76.3] | 65.5 [45.67 to 82.06] | 0 [0 to 11.22]
  HIV ENV ConA1 gp140 (Clade A) IgA Ab at W16: number analyzed (Participants) | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV ConA1 gp140 (Clade A) IgA Ab at W16 | 30.0 [16.56 to 46.53] |  |  |  |  |  |  |
  HIV ENV ConA1 gp140 (Clade A) IgA Ab at W28: number analyzed (Participants) | 39 | 31 | 36 | 35 | 34 | 38 | 37 | 38
  HIV ENV ConA1 gp140 (Clade A) IgA Ab at W28 | 46.2 [30.09 to 62.82] | 51.6 [33.06 to 69.85] | 41.7 [25.51 to 59.24] | 59.24 [31.38 to 66.01] | 47.1 [29.78 to 64.87] | 36.8 [21.81 to 54.01] | 62.2 [44.76 to 77.54] | 0 [0 to 9.25]
  HIV ENV 00MSA gp140 (Clade A) IgA Ab at W16: number analyzed (Participants) | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV 00MSA gp140 (Clade A) IgA Ab at W16 | 45.0 [29.26 to 61.51] |  |  |  |  |  |  |
  HIV ENV 00MSA gp140 (Clade A) IgA Ab at W28: number analyzed (Participants) | 39 | 31 | 36 | 35 | 34 | 38 | 37 | 38
  HIV ENV 00MSA gp140 (Clade A) IgA Ab at W28 | 56.4 [39.62 to 72.19] | 64.5 [45.37 to 80.77] | 41.7 [25.51 to 59.24] | 51.4 [33.99 to 68.62] | 52.9 [35.13 to 70.22] | 47.4 [30.98 to 64.18] | 48.6 [31.92 to 65.6] | 0 [0 to 9.25]
  HIV ENV gp41 IgA Ab at W16: number analyzed (Participants) | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HIV ENV gp41 IgA Ab at W16 | 10.0 [2.79 to 23.66] |  |  |  |  |  |  |
  HIV ENV gp41 IgA Ab at W28: number analyzed (Participants) | 39 | 31 | 36 | 35 | 34 | 38 | 37 | 38
  HIV ENV gp41 IgA Ab at W28 | 48.7 [32.42 to 65.22] | 29.0 [14.22 to 48.04] | 11.1 [3.11 to 26.06] | 42.9 [26.32 to 60.65] | 32.4 [17.39 to 50.53] | 7.9 [1.66 to 21.38] | 37.8 [22.46 to 55.24] | 2.6 [0.07 to 13.81]
  HIV ENV gp41 IgA Ab at W52: number analyzed (Participants) | 35 | 25 | 31 | 26 | 26 | 32 | 29 | 32
  HIV ENV gp41 IgA Ab at W52 | 48.6 [31.38 to 66.01] | 36.0 [17.97 to 57.48] | 9.7 [2.04 to 25.75] | 53.8 [33.37 to 73.41] | 46.2 [26.59 to 66.63] | 12.5 [3.51 to 28.99] | 58.6 [38.94 to 76.48] | 0 [0 to 10.89]
  Clade A (51802) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade A (51802) IgG-t Ab at W16 | 72.7 [57.21 to 85.04] |  |  |  |  |  |  |
  Clade A (51802) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade A (51802) IgG-t Ab at W28 | 91.3 [79.21 to 97.58] | 94.3 [80.84 to 99.3] | 88.4 [74.92 to 96.11] | 87.5 [73.2 to 95.81] | 85.7 [69.74 to 95.19] | 94.7 [82.25 to 99.36] | 85.7 [71.46 to 94.57] | 0 [0 to 8.81]
  Clade A (51802) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade A (51802) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 87.2 [72.57 to 95.7] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 86.8 [71.91 to 95.59] | 90.9 [75.67 to 98.08] | 5.6 [0.68 to 18.66]
  Clade A (51802) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade A (51802) IgG-t Ab at W78 | 79.5 [63.54 to 90.7] | 81.8 [64.54 to 93.02] |  |  |  |  |  |
  Clade A (51802) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade A (51802) IgG-t Ab at W96 | 68.4 [51.35 to 82.5] | 74.2 [55.39 to 88.14] |  |  |  |  |  |
  Clade AE (254008) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (254008) IgG-t Ab at W16 | 84.1 [69.93 to 93.36] |  |  |  |  |  |  |
  Clade AE (254008) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade AE (254008) IgG-t Ab at W28 | 89.1 [76.43 to 96.38] | 97.1 [85.08 to 99.93] | 88.4 [74.92 to 96.11] | 85.0 [70.16 to 94.29] | 85.7 [69.74 to 95.19] | 97.4 [86.19 to 99.93] | 88.1 [74.37 to 96.02] | 0 [0 to 8.81]
  Clade AE (254008) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade AE (254008) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 87.2 [72.57 to 95.7] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 92.1 [78.62 to 98.34] | 93.9 [79.77 to 99.26] | 0 [0 to 9.74]
  Clade AE (254008) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (254008) IgG-t Ab at W78 | 97.4 [86.52 to 99.94] | 97.0 [84.24 to 99.92] |  |  |  |  |  |
  Clade AE (254008) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (254008) IgG-t Ab at W96 | 94.7 [82.25 to 99.36] | 90.3 [74.25 to 97.96] |  |  |  |  |  |
  Clade AE (A244) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (A244) IgG-t Ab at W16 | 75.0 [59.66 to 86.81] |  |  |  |  |  |  |
  Clade AE (A244) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade AE (A244) IgG-t Ab at W28 | 91.3 [79.21 to 97.58] | 91.4 [76.94 to 98.2] | 81.4 [66.6 to 91.61] | 90.0 [76.34 to 97.21] | 85.7 [69.74 to 95.19] | 94.7 [82.25 to 99.36] | 88.1 [74.37 to 96.02] | 0 [0 to 8.81]
  Clade AE (A244) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade AE (A244) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 89.7 [75.78 to 97.13] | 91.2 [76.32 to 98.14] | 97.0 [84.24 to 99.92] | 89.5 [75.2 to 97.06] | 90.9 [75.67 to 98.08] | 0 [0 to 9.74]
  Clade AE (A244) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (A244) IgG-t Ab at W78 | 84.6 [69.47 to 94.14] | 84.8 [68.1 to 94.89] |  |  |  |  |  |
  Clade AE (A244) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (A244) IgG-t Ab at W96 | 71.1 [54.1 to 84.58] | 71.0 [51.96 to 85.78] |  |  |  |  |  |
  Clade B (B.6240) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (B.6240) IgG-t Ab at W16 | 86.4 [72.65 to 94.83] |  |  |  |  |  |  |
  Clade B (B.6240) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade B (B.6240) IgG-t Ab at W28 | 95.7 [85.16 to 99.47] | 97.1 [85.08 to 99.93] | 97.7 [87.71 to 99.94] | 92.5 [79.61 to 98.43] | 85.7 [69.74 to 95.19] | 97.4 [86.19 to 99.93] | 90.5 [77.38 to 97.34] | 0 [0 to 8.81]
  Clade B (B.6240) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 43 | 45
  Clade B (B.6240) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 92.3 [79.13 to 98.38] | 94.1 [80.32 to 99.28] | 100.0 [89.42 to 100.0] | 97.4 [86.19 to 99.93] | 93.9 [79.77 to 99.26] | 0 [0 to 9.74]
  Clade B (B.6240) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (B.6240) IgG-t Ab at W78 | 84.6 [69.47 to 94.14] | 93.9 [79.77 to 99.26] |  |  |  |  |  |
  Clade B (B.6240) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (B.6240) IgG-t Ab at W96 | 86.8 [71.91 to 95.59] | 93.5 [78.58 to 99.21] |  |  |  |  |  |
  Clade B (BORI) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (BORI) IgG-t Ab at W16 | 95.5 [84.53 to 99.44] |  |  |  |  |  |  |
  Clade B (BORI) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade B (BORI) IgG-t Ab at W28 | 95.7 [85.16 to 99.47] | 97.1 [85.08 to 99.93] | 93.0 [80.94 to 98.54] | 90.0 [76.34 to 97.21] | 88.6 [73.26 to 96.8] | 97.4 [86.19 to 99.93] | 90.5 [77.38 to 97.34] | 0 [0 to 8.81]
  Clade B (BORI) IgG-t Ab at Week 52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade B (BORI) IgG-t Ab at Week 52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 97.4 [86.52 to 99.94] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 97.4 [86.19 to 99.93] | 93.9 [79.77 to 99.26] | 0 [0 to 9.74]
  Clade B (BORI) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (BORI) IgG-t Ab at W78 | 84.6 [69.47 to 94.14] | 84.8 [68.1 to 94.89] |  |  |  |  |  |
  Clade B (BORI) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (BORI) IgG-t Ab at W96 | 73.7 [56.9 to 86.6] | 74.2 [55.39 to 88.14] |  |  |  |  |  |
  Clade B (TT31P) gp120 IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (TT31P) gp120 IgG-t Ab at W16 | 90.9 [78.33 to 97.47] |  |  |  |  |  |  |
  Clade B (TT31P) gp120 IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade B (TT31P) gp120 IgG-t Ab at W28 | 95.7 [85.16 to 99.47] | 91.4 [76.94 to 98.2] | 90.7 [77.86 to 97.41] | 92.5 [79.61 to 98.43] | 88.6 [73.26 to 96.8] | 100.0 [90.75 to 100.0] | 88.1 [74.37 to 96.02] | 0 [0 to 8.81]
  Clade B (TT31P) gp120 IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade B (TT31P) gp120 IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 94.9 [82.68 to 99.37] | 94.1 [80.32 to 99.28] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 90.9 [75.67 to 98.08] | 0 [0 to 9.74]
  Clade B (TT31P) gp120 IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (TT31P) gp120 IgG-t Ab at W78 | 87.2 [72.57 to 95.7] | 93.9 [79.77 to 99.26] |  |  |  |  |  |
  Clade B (TT31P) gp120 IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (TT31P) gp120 IgG-t Ab at W96 | 86.8 [71.91 to 95.59] | 87.1 [70.17 to 96.37] |  |  |  |  |  |
  Clade BC (CNE20) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade BC (CNE20) IgG-t Ab at W16 | 90.9 [78.33 to 97.47] |  |  |  |  |  |  |
  Clade BC (CNE20) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade BC (CNE20) IgG-t Ab at W28 | 93.5 [82.1 to 98.63] | 94.3 [80.84 to 99.3] | 90.7 [77.86 to 97.41] | 90.0 [76.34 to 97.21] | 88.6 [73.26 to 96.8] | 97.4 [86.19 to 99.93] | 92.9 [80.52 to 98.5] | 0 [0 to 8.81]
  Clade BC (CNE20) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade BC (CNE20) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 97.4 [86.52 to 99.94] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 94.7 [82.25 to 99.36] | 93.9 [79.77 to 99.26] | 0 [0 to 9.74]
  Clade BC (CNE20) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade BC (CNE20) IgG-t Ab at W78 | 84.6 [69.47 to 94.14] | 93.9 [79.77 to 99.26] |  |  |  |  |  |
  Clade BC (CNE20) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade BC (CNE20) IgG-t Ab at W96 | 78.9 [62.68 to 90.45] | 87.1 [70.17 to 96.37] |  |  |  |  |  |
  Clade BC(BJOX002) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade BC(BJOX002) IgG-t Ab at W16 | 75.0 [59.66 to 86.81] |  |  |  |  |  |  |
  Clade BC(BJOX002) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade BC(BJOX002) IgG-t Ab at W28 | 87.0 [73.74 to 95.06] | 94.3 [80.84 to 99.3] | 88.4 [74.92 to 96.11] | 85.0 [70.16 to 94.29] | 82.9 [66.35 to 93.44] | 89.5 [75.2 to 97.06] | 90.5 [77.38 to 97.34] | 0 [0 to 8.81]
  Clade BC(BJOX002) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade BC(BJOX002) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 89.7 [75.78 to 97.13] | 97.1 [84.67 to 99.93] | 97.0 [84.24 to 99.92] | 94.7 [82.25 to 99.36] | 93.9 [79.77 to 99.26] | 0 [0 to 9.74]
  Clade BC(BJOX002) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade BC(BJOX002) IgG-t Ab at W78 | 74.4 [57.87 to 86.96] | 75.8 [57.74 to 88.91] |  |  |  |  |  |
  Clade BC(BJOX002) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade BC(BJOX002) IgG-t Ab at W96 | 68.4 [51.35 to 82.5] | 74.2 [55.39 to 88.14] |  |  |  |  |  |
  Clade C(1086C_D7) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C(1086C_D7) IgG-t Ab at W16 | 97.7 [87.98 to 99.94] |  |  |  |  |  |  |
  Clade C(1086C_D7) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade C(1086C_D7) IgG-t Ab at W28 | 100.0 [92.29 to 100.0] | 97.1 [85.08 to 99.93] | 100.0 [91.78 to 100.0] | 97.5 [86.84 to 99.94] | 88.6 [73.26 to 96.8] | 100.0 [90.75 to 100.0] | 90.75 [83.84 to 99.42] | 0 [0 to 8.81]
  Clade C(1086C_D7) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade C(1086C_D7) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 100.0 [90.97 to 100.0] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 97.0 [84.24 to 99.92] | 0 [0 to 9.74]
  Clade C(1086C_D7) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C(1086C_D7) IgG-t Ab at W78 | 100.0 [90.97 to 100.0] | 100.0 [89.42 to 100.0] |  |  |  |  |  |
  Clade C(1086C_D7) IgG-t Ab at Week 96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C(1086C_D7) IgG-t Ab at Week 96 | 97.4 [86.19 to 99.93] | 96.8 [83.3 to 99.92] |  |  |  |  |  |
  B Clade M (Con 6) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  B Clade M (Con 6) IgG-t Ab at W16 | 97.7 [87.98 to 99.94] |  |  |  |  |  |  |
  B Clade M (Con 6) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  B Clade M (Con 6) IgG-t Ab at W28 | 97.8 [88.47 to 99.94] | 97.1 [85.08 to 99.93] | 97.7 [87.71 to 99.94] | 92.5 [79.61 to 98.43] | 88.6 [73.26 to 96.8] | 100.0 [90.75 to 100.0] | 92.9 [80.52 to 98.5] | 0 [0 to 8.81]
  B Clade M (Con 6) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  B Clade M (Con 6) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 97.4 [86.52 to 99.94] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 97.0 [84.24 to 99.92] | 0 [0 to 9.74]
  B Clade M (Con 6) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  B Clade M (Con 6) IgG-t Ab at W78 | 97.4 [86.52 to 99.94] | 97.0 [84.24 to 99.92] |  |  |  |  |  |
  B Clade M (Con 6) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  B Clade M (Con 6) IgG-t Ab at W96 | 92.1 [78.62 to 98.34] | 93.5 [78.58 to 99.21] |  |  |  |  |  |
  Clade B (SC42261) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (SC42261) IgG-t Ab at W16 | 95.5 [84.53 to 99.44] |  |  |  |  |  |  |
  Clade B (SC42261) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade B (SC42261) IgG-t Ab at W28 | 97.8 [88.47 to 99.94] | 97.1 [85.08 to 99.93] | 100.0 [91.78 to 100.0] | 95.0 [83.08 to 99.39] | 88.6 [73.26 to 96.8] | 100.0 [90.75 to 100.0] | 95.2 [83.84 to 99.42] | 0 [0 to 8.81]
  Clade B (SC42261) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade B (SC42261) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 100.0 [90.97 to 100.0] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 97.0 [84.24 to 99.92] | 0 [0 to 9.74]
  Clade B (SC42261) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (SC42261) IgG-t Ab at W78 | 92.3 [79.13 to 98.38] | 97.0 [84.24 to 99.92] |  |  |  |  |  |
  Clade B (SC42261) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (SC42261) IgG-t Ab at W96 | 92.1 [78.62 to 98.34] | 93.5 [78.58 to 99.21] |  |  |  |  |  |
  Clade C (CH505TF) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (CH505TF) IgG-t Ab at W16 | 88.6 [75.44 to 96.21] |  |  |  |  |  |  |
  Clade C (CH505TF) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade C (CH505TF) IgG-t Ab at W28 | 93.5 [82.1 to 98.63] | 97.1 [85.08 to 99.93] | 93.0 [80.94 to 98.54] | 92.5 [79.61 to 98.43] | 85.7 [69.74 to 95.19] | 97.4 [86.19 to 99.93] | 95.2 [83.84 to 99.42] | 0 [0 to 8.81]
  Clade C (CH505TF) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade C (CH505TF) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 92.3 [79.13 to 98.38] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 97.0 [84.24 to 99.92] | 0 [0 to 9.74]
  Clade C (CH505TF) IgG-t Ab at W78: number analyzed (Participants) | 38 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (CH505TF) IgG-t Ab at W78 | 84.2 [68.75 to 93.98] | 90.9 [75.67 to 98.08] |  |  |  |  |  |
  Clade C (CH505TF) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (CH505TF) IgG-t Ab at W96 | 81.6 [65.67 to 92.26] | 77.4 [58.9 to 90.41] |  |  |  |  |  |
  C Clade A (9004S) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade A (9004S) IgG-t Ab at W16 | 84.1 [69.93 to 93.36] |  |  |  |  |  |  |
  C Clade A (9004S) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  C Clade A (9004S) IgG-t Ab at W28 | 91.3 [79.21 to 97.58] | 94.3 [80.84 to 99.3] | 90.7 [77.86 to 97.41] | 90.0 [76.34 to 97.21] | 85.7 [69.74 to 95.19] | 97.4 [86.19 to 99.93] | 88.1 [74.37 to 96.02] | 0 [0 to 8.81]
  C Clade A (9004S) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  C Clade A (9004S) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 94.9 [82.68 to 99.37] | 100.0 [89.72 to 100.0] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 93.9 [79.77 to 99.26] | 0 [0 to 9.74]
  C Clade A (9004S) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade A (9004S) IgG-t Ab at W78 | 87.2 [72.57 to 95.7] | 84.8 [68.1 to 94.89] |  |  |  |  |  |
  C Clade A (9004S) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade A (9004S) IgG-t Ab at W96 | 86.8 [71.91 to 95.59] | 87.1 [70.17 to 96.37] |  |  |  |  |  |
  C Clade B (RHPA) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade B (RHPA) IgG-t Ab at W16 | 97.7 [87.98 to 99.94] |  |  |  |  |  |  |
  C Clade B (RHPA) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  C Clade B (RHPA) IgG-t Ab at W28 | 97.8 [88.47 to 99.94] | 97.1 [85.08 to 99.93] | 100.0 [91.78 to 100.0] | 92.5 [79.61 to 98.43] | 88.6 [73.26 to 96.8] | 100.0 [90.75 to 100.0] | 95.2 [83.84 to 99.42] | 0 [0 to 8.81]
  C Clade B (RHPA) IgG-t Ab at Week 52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  C Clade B (RHPA) IgG-t Ab at Week 52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 100.0 [90.97 to 100.0] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 97.0 [84.24 to 99.92] | 2.8 [0.07 to 14.53]
  C Clade B (RHPA) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade B (RHPA) IgG-t Ab at W78 | 92.3 [79.13 to 98.38] | 97.0 [84.24 to 99.92] |  |  |  |  |  |
  C Clade B (RHPA) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade B (RHPA) IgG-t Ab at W96 | 92.1 [78.62 to 98.34] | 93.5 [78.58 to 99.21] |  |  |  |  |  |
  C Clade B (WITO) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade B (WITO) IgG-t Ab at W16 | 93.2 [81.34 to 98.57] |  |  |  |  |  |  |
  C Clade B (WITO) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  C Clade B (WITO) IgG-t Ab at W28 | 97.8 [88.47 to 99.94] | 97.1 [85.08 to 99.93] | 97.7 [87.71 to 99.94] | 92.5 [79.61 to 98.43] | 88.6 [73.26 to 96.8] | 100.0 [90.75 to 100.0] | 95.2 [83.84 to 99.42] | 0 [0 to 8.81]
  C Clade B (WITO) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  C Clade B (WITO) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 97.4 [86.52 to 99.94] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 97.0 [84.24 to 99.92] | 0 [0 to 9.74]
  C Clade B (WITO) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade B (WITO) IgG-t Ab at W78 | 87.2 [72.57 to 95.7] | 97.0 [84.24 to 99.92] |  |  |  |  |  |
  C Clade B (WITO) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade B (WITO) IgG-t Ab at W96 | 92.1 [78.62 to 98.34] | 93.5 [78.58 to 99.21] |  |  |  |  |  |
  C Clade C (1086C) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade C (1086C) IgG-t Ab at W16 | 97.7 [87.98 to 99.94] |  |  |  |  |  |  |
  C Clade C (1086C) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  C Clade C (1086C) IgG-t Ab at W28 | 100.0 [92.29 to 100.0] | 97.1 [85.08 to 99.93] | 100.0 [91.78 to 100.0] | 97.5 [86.84 to 99.94] | 88.6 [73.26 to 96.8] | 100.0 [90.75 to 100.0] | 97.6 [87.43 to 99.94] | 2.5 [0.06 to 13.16]
  C Clade C (1086C) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  C Clade C (1086C) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 100.0 [90.97 to 100.0] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 97.0 [84.24 to 99.92] | 0 [0 to 9.74]
  C Clade C (1086C) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade C (1086C) IgG-t Ab at W78 | 100.0 [90.97 to 100.0] | 100.0 [89.42 to 100.0] |  |  |  |  |  |
  C Clade C (1086C) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade C (1086C) IgG-t Ab at W96 | 100.0 [90.75 to 100.0] | 96.8 [83.3 to 99.92] |  |  |  |  |  |
  C Clade C (BF1266) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade C (BF1266) IgG-t Ab at W16 | 93.2 [81.34 to 98.57] |  |  |  |  |  |  |
  C Clade C (BF1266) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  C Clade C (BF1266) IgG-t Ab at W28 | 95.7 [85.16 to 99.47] | 97.1 [85.08 to 99.93] | 97.7 [87.71 to 99.94] | 92.5 [79.61 to 98.43] | 88.6 [73.26 to 96.8] | 100.0 [90.75 to 100.0] | 92.9 [80.52 to 98.5] | 2.5 [0.06 to 13.16]
  C Clade C (BF1266) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  C Clade C (BF1266) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 100.0 [90.97 to 100.0] | 100.0 [89.72 to 100.0] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 97.0 [84.24 to 99.92] | 2.8 [0.07 to 14.53]
  C Clade C (BF1266) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade C (BF1266) IgG-t Ab at W78 | 92.3 [79.13 to 98.38] | 100.0 [89.42 to 100.0] |  |  |  |  |  |
  C Clade C (BF1266) IgG-t Ab at Week 96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  C Clade C (BF1266) IgG-t Ab at Week 96 | 92.1 [78.62 to 98.34] | 93.5 [78.58 to 99.21] |  |  |  |  |  |
  CF Clade AE (conAE) IgG-t Ab at 16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CF Clade AE (conAE) IgG-t Ab at 16 | 88.6 [75.44 to 96.21] |  |  |  |  |  |  |
  CF Clade AE (conAE) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  CF Clade AE (conAE) IgG-t Ab at W28 | 95.7 [85.16 to 99.47] | 97.1 [85.08 to 99.93] | 93.0 [80.94 to 98.54] | 90.0 [76.34 to 97.21] | 85.7 [69.74 to 95.19] | 97.4 [86.19 to 99.93] | 95.2 [83.84 to 99.42] | 0 [0 to 8.81]
  CF Clade AE (conAE) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  CF Clade AE (conAE) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 92.3 [79.13 to 98.38] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 97.4 [86.19 to 99.93] | 97.0 [84.24 to 99.92] | 0 [0 to 9.74]
  CF Clade AE (conAE) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  CF Clade AE (conAE) IgG-t Ab at W78 | 92.3 [79.13 to 98.38] | 97.0 [84.24 to 99.92] |  |  |  |  |  |
  CF Clade AE (conAE) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  CF Clade AE (conAE) IgG-t Ab at W96 | 84.2 [68.75 to 93.98] | 87.1 [70.17 to 96.37] |  |  |  |  |  |
  CFI Clade M(Con S) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFI Clade M(Con S) IgG-t Ab at W16 | 97.7 [87.98 to 99.94] |  |  |  |  |  |  |
  CFI Clade M(Con S) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  CFI Clade M(Con S) IgG-t Ab at W28 | 100.0 [92.29 to 100.0] | 97.1 [85.08 to 99.93] | 100.0 [91.78 to 100.0] | 97.5 [86.84 to 99.94] | 88.6 [73.26 to 96.8] | 100.0 [90.75 to 100.0] | 97.6 [87.43 to 99.94] | 0 [0 to 8.81]
  CFI Clade M(Con S) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  CFI Clade M(Con S) IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 100.0 [90.97 to 100.0] | 97.1 [84.67 to 99.93] | 100.0 [89.42 to 100.0] | 100.0 [90.75 to 100.0] | 100.0 [89.42 to 100.0] | 0 [0 to 9.74]
  CFI Clade M(Con S) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  CFI Clade M(Con S) IgG-t Ab at W78 | 100.0 [90.97 to 100.0] | 100.0 [89.42 to 100.0] |  |  |  |  |  |
  CFI Clade M(Con S) IgG-t Ab at Week 96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  CFI Clade M(Con S) IgG-t Ab at Week 96 | 100.0 [90.75 to 100.0] | 96.8 [83.3 to 99.92] |  |  |  |  |  |
  IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  IgG-t Ab at W16 | 72.7 [57.21 to 85.04] |  |  |  |  |  |  |
  IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  IgG-t Ab at W28 | 95.7 [85.16 to 99.47] | 88.6 [73.26 to 96.8] | 79.1 [63.96 to 89.96] | 87.5 [73.2 to 95.81] | 85.7 [69.74 to 95.19] | 89.5 [75.2 to 97.06] | 90.5 [77.38 to 97.34] | 0 [0 to 8.81]
  IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  IgG-t Ab at W52 | 100.0 [90.51 to 100.0] | 100.0 [89.11 to 100.0] | 89.7 [75.78 to 97.13] | 97.1 [84.67 to 99.93] | 97.0 [84.24 to 99.92] | 92.1 [78.62 to 98.34] | 97.0 [84.24 to 99.92] | 5.6 [0.68 to 18.66]
  IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  IgG-t Ab at W78 | 87.2 [72.57 to 95.7] | 81.8 [64.54 to 93.02] |  |  |  |  |  |
  IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  IgG-t Ab at W96 | 81.6 [65.67 to 92.26] | 67.7 [48.63 to 83.32] |  |  |  |  |  |
  Clade A (191084) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade A (191084) IgG-t Ab at W16 | 47.7 [32.46 to 63.31] |  |  |  |  |  |  |
  Clade A (191084) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade A (191084) IgG-t Ab at W28 | 65.2 [49.75 to 78.65] | 45.7 [28.83 to 63.35] | 46.5 [31.18 to 62.35] | 60.0 [43.33 to 75.14] | 42.9 [26.32 to 60.65] | 47.4 [30.98 to 64.18] | 38.1 [23.57 to 54.36] | 0 [0 to 8.81]
  Clade A (191084) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade A (191084) IgG-t Ab at W52 | 81.1 [64.84 to 92.04] | 62.5 [43.69 to 78.9] | 59.0 [42.1 to 74.43] | 73.5 [55.64 to 87.12] | 75.8 [57.74 to 88.91] | 57.9 [40.82 to 73.69] | 51.5 [33.54 to 69.2] | 0 [0 to 9.74]
  Clade A (191084) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade A (191084) IgG-t Ab at W78 | 28.2 [15 to 44.87] | 18.2 [6.98 to 35.46] |  |  |  |  |  |
  Clade A (191084) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade A (191084) IgG-t Ab at W96 | 21.1 [9.55 to 37.32] | 16.1 [5.45 to 33.73] |  |  |  |  |  |
  Clade AE (C2101) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (C2101) IgG-t Ab at W16 | 47.7 [32.46 to 63.31] |  |  |  |  |  |  |
  Clade AE (C2101) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade AE (C2101) IgG-t Ab at W28 | 58.7 [43.23 to 73] | 45.7 [28.83 to 63.35] | 48.8 [33.31 to 64.54] | 62.5 [45.8 to 77.27] | 48.6 [31.38 to 66.01] | 52.6 [35.82 to 69.02] | 28.6 [15.72 to 44.58] | 0 [0 to 8.81]
  Clade AE (C2101) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade AE (C2101) IgG-t Ab at W52 | 73.0 [55.88 to 86.21] | 59.4 [40.64 to 76.3] | 61.5 [44.62 to 76.64] | 79.4 [62.1 to 91.3] | 69.7 [51.29 to 84.41] | 55.3 [38.3 to 71.38] | 36.4 [20.4 to 54.88] | 2.8 [0.07 to 14.53]
  Clade AE (C2101) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (C2101) IgG-t Ab at W78 | 28.2 [15 to 44.87] | 30.3 [15.59 to 48.71] |  |  |  |  |  |
  Clade AE (C2101) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (C2101) IgG-t Ab at W96 | 21.1 [9.55 to 37.32] | 32.3 [16.68 to 51.37] |  |  |  |  |  |
  Clade AE (CM244) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (CM244) IgG-t Ab at W16 | 47.7 [32.46 to 63.31] |  |  |  |  |  |  |
  Clade AE (CM244) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 34 | 38 | 42 | 40
  Clade AE (CM244) IgG-t Ab at W28 | 58.7 [43.23 to 73] | 37.1 [21.47 to 55.08] | 46.5 [31.18 to 62.35] | 57.5 [40.89 to 72.96] | 29.4 [15.1 to 47.48] | 42.1 [26.31 to 59.18] | 28.6 [15.72 to 44.58] | 0 [0 to 8.81]
  Clade AE (CM244) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade AE (CM244) IgG-t Ab at W52 | 83.8 [67.99 to 93.81] | 56.3 [37.66 to 73.64] | 56.4 [39.62 to 72.19] | 76.5 [58.83 to 89.25] | 57.6 [39.22 to 74.52] | 57.9 [40.82 to 73.69] | 42.4 [25.48 to 60.78] | 0 [0 to 9.74]
  Clade AE (CM244) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (CM244) IgG-t Ab at W78 | 23.1 [11.13 to 39.33] | 12.1 [3.4 to 28.2] |  |  |  |  |  |
  Clade AE (CM244) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade AE (CM244) IgG-t Ab at W96 | 21.1 [9.55 to 37.32] | 16.1 [5.45 to 33.73] |  |  |  |  |  |
  Clade B (62357.14) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (62357.14) IgG-t Ab at W16 | 22.7 [11.47 to 37.84] |  |  |  |  |  |  |
  Clade B (62357.14) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade B (62357.14) IgG-t Ab at W28 | 41.3 [27 to 56.77] | 17.1 [6.56 to 33.65] | 16.3 [6.81 to 30.7] | 37.5 [22.73 to 54.2] | 20.0 [8.44 to 36.94] | 23.7 [11.44 to 40.24] | 19.0 [8.6 to 34.12] | 0 [0 to 8.81]
  Clade B (62357.14) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade B (62357.14) IgG-t Ab at W52 | 59.5 [42.1 to 75.25] | 34.4 [18.57 to 53.19] | 20.5 [9.3 to 36.46] | 61.8 [43.56 to 77.83] | 45.5 [28.11 to 63.65] | 26.3 [13.4 to 43.1] | 36.4 [20.4 to 54.88] | 0 [0 to 9.74]
  Clade B (62357.14) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (62357.14) IgG-t Ab at W78 | 20.5 [9.3 to 36.46] | 9.1 [1.92 to 24.33] |  |  |  |  |  |
  Clade B (62357.14) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (62357.14) IgG-t Ab at W96 | 10.5 [2.94 to 24.8] | 12.9 [3.63 to 29.83] |  |  |  |  |  |
  Clade B (CaseA) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (CaseA) IgG-t Ab at W16 | 59.1 [43.25 to 73.66] |  |  |  |  |  |  |
  Clade B (CaseA) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade B (CaseA) IgG-t Ab at W28 | 67.4 [51.98 to 80.47] | 51.4 [33.99 to 68.62] | 62.8 [46.73 to 77.02] | 65.0 [48.32 to 79.37] | 42.9 [26.32 to 60.65] | 63.2 [45.99 to 78.19] | 45.2 [29.85 to 61.33] | 0 [0 to 8.81]
  Clade B (CaseA) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade B (CaseA) IgG-t Ab at W52 | 86.5 [71.23 to 95.46] | 75.0 [56.6 to 88.54] | 71.8 [55.13 to 85] | 70.6 [52.52 to 84.9] | 81.8 [64.54 to 93.02] | 71.1 [54.1 to 84.58] | 60.6 [42.14 to 77.09] | 13.9 [4.67 to 29.5]
  Clade B (CaseA) IgG-t Ab at W78: number analyzed (Participants) | 38 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (CaseA) IgG-t Ab at W78 | 42.1 [26.31 to 59.18] | 30.3 [15.59 to 48.71] |  |  |  |  |  |
  Clade B (CaseA) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (CaseA) IgG-t Ab at W96 | 28.9 [15.42 to 45.9] | 29.0 [14.22 to 48.04] |  |  |  |  |  |
  Clade B (RHPA4259) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (RHPA4259) IgG-t Ab at W16 | 50.0 [34.56 to 65.44] |  |  |  |  |  |  |
  Clade B (RHPA4259) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 34 | 38 | 42 | 40
  Clade B (RHPA4259) IgG-t Ab at W28 | 69.6 [54.25 to 82.26] | 48.6 [31.38 to 66.01] | 51.2 [35.46 to 66.69] | 60.0 [43.33 to 75.14] | 47.1 [29.78 to 64.87] | 50.0 [33.38 to 66.62] | 35.7 [21.55 to 51.97] | 0 [0 to 8.81]
  Clade B (RHPA4259) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade B (RHPA4259) IgG-t Ab at W52 | 83.8 [67.99 to 93.81] | 59.4 [40.64 to 76.3] | 59.0 [42.1 to 74.43] | 67.6 [49.47 to 82.61] | 75.8 [57.74 to 88.91] | 57.9 [40.82 to 73.69] | 48.5 [30.8 to 66.46] | 0 [0 to 9.74]
  Clade B (RHPA4259) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (RHPA4259) IgG-t Ab at W78 | 33.3 [19.09 to 50.22] | 18.2 [6.98 to 35.46] |  |  |  |  |  |
  Clade B (RHPA4259) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (RHPA4259) IgG-t Ab at W96 | 28.9 [15.42 to 45.9] | 22.6 [9.59 to 41.1] |  |  |  |  |  |
  Clade B (TT31P) gp70 IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (TT31P) gp70 IgG-t Ab at W16 | 59.1 [43.25 to 73.66] |  |  |  |  |  |  |
  Clade B (TT31P) gp70 IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade B (TT31P) gp70 IgG-t Ab at W28 | 69.6 [54.25 to 82.26] | 45.7 [28.83 to 63.35] | 51.2 [35.46 to 66.69] | 62.5 [45.8 to 77.27] | 37.1 [21.47 to 55.08] | 50.0 [33.38 to 66.62] | 50.0 [34.19 to 65.81] | 0 [0 to 8.81]
  Clade B (TT31P) gp70 IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade B (TT31P) gp70 IgG-t Ab at W52 | 86.5 [71.23 to 95.46] | 62.5 [43.69 to 78.9] | 66.7 [49.78 to 80.91] | 73.5 [55.64 to 87.12] | 75.8 [57.74 to 88.91] | 57.9 [40.82 to 73.69] | 57.6 [39.22 to 74.52] | 2.8 [0.07 to 14.53]
  Clade B (TT31P) gp70 IgG-t Ab at W78: number analyzed (Participants) | 38 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (TT31P) gp70 IgG-t Ab at W78 | 36.8 [21.81 to 54.01] | 24.2 [11.09 to 42.26] |  |  |  |  |  |
  Clade B (TT31P) gp70 IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B (TT31P) gp70 IgG-t Ab at W96 | 31.6 [17.5 to 48.65] | 22.6 [9.59 to 41.1] |  |  |  |  |  |
  Clade B(700010058) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B(700010058) IgG-t Ab at W16 | 50.0 [34.56 to 65.44] |  |  |  |  |  |  |
  Clade B(700010058) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade B(700010058) IgG-t Ab at W28 | 60.9 [45.37 to 74.91] | 45.7 [28.83 to 63.35] | 53.5 [37.65 to 68.82] | 62.5 [45.8 to 77.27] | 37.1 [21.47 to 55.08] | 50.0 [33.38 to 66.62] | 26.2 [13.86 to 42.04] | 0 [0 to 8.81]
  Clade B(700010058) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade B(700010058) IgG-t Ab at W52 | 64.9 [47.46 to 79.79] | 62.5 [43.69 to 78.9] | 64.1 [47.18 to 78.8] | 70.6 [52.52 to 84.9] | 66.7 [48.17 to 82.04] | 57.9 [40.82 to 73.69] | 33.3 [17.96 to 51.83] | 0 [0 to 9.74]
  Clade B(700010058) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B(700010058) IgG-t Ab at W78 | 28.2 [15 to 44.87] | 30.3 [15.59 to 48.71] |  |  |  |  |  |
  Clade B(700010058) IgG-t Ab at W96: number analyzed (Participants) | 37 | 30 | 0 | 0 | 0 | 0 | 0 | 0
  Clade B(700010058) IgG-t Ab at W96 | 27.0 [13.79 to 44.12] | 23.3 [9.93 to 42.28] |  |  |  |  |  |
  Clade BC (BJOX) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade BC (BJOX) IgG-t Ab at W16 | 52.3 [36.69 to 67.54] |  |  |  |  |  |  |
  Clade BC (BJOX) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade BC (BJOX) IgG-t Ab at W28 | 67.4 [51.98 to 80.47] | 48.6 [31.38 to 66.01] | 55.8 [39.88 to 70.92] | 62.5 [45.8 to 77.27] | 40.0 [23.87 to 57.89] | 47.4 [30.98 to 64.18] | 35.7 [21.55 to 51.97] | 0 [0 to 8.81]
  Clade BC (BJOX) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade BC (BJOX) IgG-t Ab at W52 | 81.1 [64.84 to 92.04] | 62.5 [43.69 to 78.9] | 66.7 [49.78 to 80.91] | 70.6 [52.52 to 84.9] | 66.7 [48.17 to 82.04] | 60.5 [43.39 to 75.96] | 54.5 [36.35 to 71.89] | 2.8 [0.07 to 14.53]
  Clade BC (BJOX) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade BC (BJOX) IgG-t Ab at W78 | 23.1 [11.13 to 39.33] | 18.2 [6.98 to 35.46] |  |  |  |  |  |
  Clade BC (BJOX) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade BC (BJOX) IgG-t Ab at W96 | 21.1 [9.55 to 37.32] | 22.6 [9.59 to 41.1] |  |  |  |  |  |
  Clade C (96ZM651) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (96ZM651) IgG-t Ab at W16 | 13.6 [5.17 to 27.35] |  |  |  |  |  |  |
  Clade C (96ZM651) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade C (96ZM651) IgG-t Ab at W28 | 28.3 [15.99 to 43.46] | 17.1 [6.56 to 33.65] | 4.7 [0.57 to 15.81] | 32.5 [18.57 to 49.13] | 20.0 [8.44 to 36.94] | 18.4 [7.74 to 34.33] | 14.3 [5.43 to 28.54] | 0 [0 to 8.81]
  Clade C (96ZM651) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade C (96ZM651) IgG-t Ab at W52 | 54.1 [36.92 to 70.51] | 40.6 [23.7 to 59.36] | 20.5 [9.3 to 36.46] | 61.8 [43.56 to 77.83] | 36.4 [20.4 to 54.88] | 36.8 [21.81 to 54.01] | 30.3 [15.59 to 48.71] | 2.8 [0.07 to 14.53]
  Clade C (96ZM651) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (96ZM651) IgG-t Ab at W78 | 10.3 [2.87 to 24.22] | 9.1 [1.92 to 24.33] |  |  |  |  |  |
  Clade C (96ZM651) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (96ZM651) IgG-t Ab at W96 | 10.5 [2.94 to 24.8] | 6.5 [0.79 to 21.42] |  |  |  |  |  |
  Clade C (BF1266) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (BF1266) IgG-t Ab at W16 | 43.2 [28.35 to 58.97] |  |  |  |  |  |  |
  Clade C (BF1266) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade C (BF1266) IgG-t Ab at W28 | 58.7 [43.23 to 73] | 31.4 [16.85 to 49.29] | 30.2 [17.18 to 46.13] | 50.0 [33.8 to 66.2] | 34.3 [19.13 to 52.21] | 34.2 [19.63 to 51.35] | 31.0 [17.62 to 47.09] | 0 [0 to 8.81]
  Clade C (BF1266) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade C (BF1266) IgG-t Ab at W52 | 78.4 [61.79 to 90.17] | 43.8 [26.36 to 62.34] | 43.6 [27.81 to 60.38] | 70.6 [52.52 to 84.9] | 51.5 [33.54 to 69.2] | 42.1 [26.31 to 59.18] | 48.5 [30.8 to 66.46] | 0 [0 to 9.74]
  Clade C (BF1266) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (BF1266) IgG-t Ab at W78 | 17.9 [7.54 to 33.53] | 18.2 [6.98 to 35.46] |  |  |  |  |  |
  Clade C (BF1266) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (BF1266) IgG-t Ab at W96 | 18.4 [7.74 to 34.33] | 22.6 [9.59 to 41.1] |  |  |  |  |  |
  Clade C (CAP210) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (CAP210) IgG-t Ab at W16 | 34.1 [20.49 to 49.92] |  |  |  |  |  |  |
  Clade C (CAP210) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade C (CAP210) IgG-t Ab at W28 | 47.8 [32.89 to 63.05] | 42.9 [26.32 to 60.65] | 32.6 [19.08 to 48.54] | 50.0 [33.8 to 66.2] | 25.7 [12.49 to 43.26] | 21.1 [9.55 to 37.32] | 26.2 [13.86 to 42.04] | 0 [0 to 8.81]
  Clade C (CAP210) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade C (CAP210) IgG-t Ab at W52 | 67.6 [50.21 to 81.99] | 53.1 [34.74 to 70.91] | 43.6 [27.81 to 60.38] | 67.6 [49.47 to 82.61] | 51.5 [33.54 to 69.2] | 39.5 [24.04 to 56.61] | 48.5 [30.8 to 66.46] | 0 [0 to 9.74]
  Clade C (CAP210) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (CAP210) IgG-t Ab at W78 | 25.6 [13.04 to 42.13] | 18.2 [6.98 to 35.46] |  |  |  |  |  |
  Clade C (CAP210) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (CAP210) IgG-t Ab at W96 | 21.1 [9.55 to 37.32] | 16.1 [5.45 to 33.73] |  |  |  |  |  |
  Clade C(Ce1086) IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C(Ce1086) IgG-t Ab at W16 | 47.7 [32.46 to 63.31] |  |  |  |  |  |  |
  Clade C(Ce1086) IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 34 | 38 | 42 | 40
  Clade C(Ce1086) IgG-t Ab at W28 | 65.2 [49.75 to 78.65] | 48.6 [31.38 to 66.01] | 55.8 [39.88 to 70.92] | 60.0 [43.33 to 75.14] | 41.2 [24.65 to 59.3] | 50.0 [33.38 to 66.62] | 35.7 [21.55 to 51.97] | 0 [0 to 8.81]
  Clade C(Ce1086) IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade C(Ce1086) IgG-t Ab at W52 | 81.1 [64.84 to 92.04] | 65.6 [46.81 to 81.43] | 64.1 [47.18 to 78.8] | 85.3 [68.94 to 95.05] | 72.7 [54.48 to 86.7] | 68.4 [51.35 to 82.5] | 54.5 [36.35 to 71.89] | 0 [0 to 9.74]
  Clade C(Ce1086) IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C(Ce1086) IgG-t Ab at W78 | 28.2 [15 to 44.87] | 18.2 [6.98 to 35.46] |  |  |  |  |  |
  Clade C(Ce1086) IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C(Ce1086) IgG-t Ab at W96 | 23.7 [11.44 to 40.24] | 22.6 [9.59 to 41.1] |  |  |  |  |  |
  Clade C(TV1.21)IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C(TV1.21)IgG-t Ab at W16 | 56.8 [41.03 to 71.65] |  |  |  |  |  |  |
  Clade C(TV1.21)IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade C(TV1.21)IgG-t Ab at W28 | 78.3 [63.64 to 89.05] | 54.3 [36.65 to 71.17] | 48.8 [33.31 to 64.54] | 62.5 [45.8 to 77.27] | 48.6 [31.38 to 66.01] | 39.5 [24.04 to 56.61] | 50.0 [34.19 to 65.81] | 0 [0 to 8.81]
  Clade C(TV1.21)IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade C(TV1.21)IgG-t Ab at W52 | 89.2 [74.58 to 96.97] | 68.8 [49.99 to 83.88] | 64.1 [47.18 to 78.8] | 79.4 [62.1 to 91.3] | 78.8 [61.09 to 91.02] | 50.0 [33.38 to 66.62] | 66.7 [48.17 to 82.04] | 2.8 [0.07 to 14.53]
  Clade C(TV1.21)IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C(TV1.21)IgG-t Ab at W78 | 38.5 [23.36 to 55.38] | 27.3 [13.3 to 45.52] |  |  |  |  |  |
  Clade C(TV1.21)IgG-t Ab at W96: number analyzed (Participants) | 37 | 30 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C(TV1.21)IgG-t Ab at W96 | 29.7 [15.87 to 46.98] | 26.7 [12.28 to 45.89] |  |  |  |  |  |
  Clade C (001428)IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (001428)IgG-t Ab at W16 | 45.5 [30.39 to 61.15] |  |  |  |  |  |  |
  Clade C (001428)IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade C (001428)IgG-t Ab at W28 | 56.5 [41.11 to 71.07] | 40.0 [23.87 to 57.89] | 37.2 [22.98 to 53.27] | 57.5 [40.89 to 72.96] | 28.6 [14.64 to 46.3] | 31.6 [17.5 to 48.65] | 35.7 [21.55 to 51.97] | 0 [0 to 8.81]
  Clade C (001428)IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade C (001428)IgG-t Ab at W52 | 81.1 [64.84 to 92.04] | 68.8 [49.99 to 83.88] | 53.8 [37.18 to 69.91] | 73.5 [55.64 to 87.12] | 66.7 [48.17 to 82.04] | 42.1 [26.31 to 59.18] | 57.6 [39.22 to 74.52] | 0 [0 to 9.74]
  Clade C (001428)IgG-t Ab at W78: number analyzed (Participants) | 40 | 32 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (001428)IgG-t Ab at W78 | 35.0 [20.63 to 51.68] | 25.0 [11.46 to 43.4] |  |  |  |  |  |
  Clade C (001428)IgG-t Ab at W96: number analyzed (Participants) | 39 | 30 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (001428)IgG-t Ab at W96 | 28.2 [15 to 44.87] | 26.7 [12.28 to 45.89] |  |  |  |  |  |
  Clade C (7060101641)IgG-t Ab at W16: number analyzed (Participants) | 44 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (7060101641)IgG-t Ab at W16 | 47.7 [32.46 to 63.31] |  |  |  |  |  |  |
  Clade C (7060101641)IgG-t Ab at W28: number analyzed (Participants) | 46 | 35 | 43 | 40 | 35 | 38 | 42 | 40
  Clade C (7060101641)IgG-t Ab at W28 | 63.0 [47.55 to 76.79] | 42.9 [26.32 to 60.65] | 48.8 [33.31 to 64.54] | 57.5 [40.89 to 72.96] | 34.3 [19.13 to 52.21] | 42.1 [26.31 to 59.18] | 33.3 [19.57 to 49.55] | 0 [0 to 8.81]
  Clade C (7060101641)IgG-t Ab at W52: number analyzed (Participants) | 37 | 32 | 39 | 34 | 33 | 38 | 33 | 36
  Clade C (7060101641)IgG-t Ab at W52 | 81.1 [64.84 to 92.04] | 62.5 [43.69 to 78.9] | 59.0 [42.1 to 74.43] | 67.6 [49.47 to 82.61] | 66.7 [48.17 to 82.04] | 44.7 [28.62 to 61.7] | 51.5 [33.54 to 69.2] | 0 [0 to 9.74]
  Clade C (7060101641)IgG-t Ab at W78: number analyzed (Participants) | 39 | 33 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (7060101641)IgG-t Ab at W78 | 38.5 [23.36 to 55.38] | 15.2 [5.11 to 31.9] |  |  |  |  |  |
  Clade C (7060101641)IgG-t Ab at W96: number analyzed (Participants) | 38 | 31 | 0 | 0 | 0 | 0 | 0 | 0
  Clade C (7060101641)IgG-t Ab at W96 | 18.4 [7.74 to 34.33] | 16.1 [5.45 to 33.73] |  |  |  |  |  |

11. Secondary Outcome: Percentage of Responders With Interferon-gamma (IFN-gamma) T Cell Responses Enzyme-linked Immunospot Assay (ELISpot)
Description: Frozen peripheral blood mononuclear cell (PBMCs) were analyzed by interferon-gamma (IFN-gamma) (ELISpot). The response was defined as post-baseline value >P95 if baseline <P95 or missing or defined as post-baseline value >3-fold increase from baseline if baseline >=P95. The threshold for ELISpot test was based on the 95th percentile (P95) from the baseline values of participants on that test in the study. Samples taken after W48 from PPI set, who missed 4th vaccine or deviated schedule were excluded. As planned, the data reported for this endpoint at specified time points only for each reported category.
Time Frame: Week 26, 50, 78 and 96
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
Number analyzed (Participants) | 47 | 39 | 45 | 44 | 43 | 38 | 43 | 46
percentage of responders
  ENV peptide pool Mos1 at Week (W) 26: number analyzed (Participants) | 47 | 39 | 44 | 44 | 43 | 38 | 43 | 46
  ENV peptide pool Mos1 at Week (W) 26 | 91.5 [79.62 to 97.63] | 79.5 [63.54 to 90.7] | 75.0 [59.66 to 86.81] | 95.5 [84.53 to 99.44] | 97.7 [87.71 to 99.94] | 92.1 [78.62 to 98.34] | 86.0 [72.07 to 94.7] | 4.3 [0.53 to 14.84]
  ENV peptide pool Mos1 at W 50: number analyzed (Participants) | 41 | 38 | 41 | 39 | 34 | 37 | 34 | 38
  ENV peptide pool Mos1 at W 50 | 87.8 [73.8 to 95.92] | 84.2 [68.75 to 93.98] | 78.0 [62.39 to 89.44] | 94.9 [82.68 to 99.37] | 97.1 [84.67 to 99.93] | 97.3 [85.84 to 99.93] | 76.5 [58.83 to 89.25] | 2.6 [0.07 to 13.81]
  ENV peptide pool Mos2 at W 26: number analyzed (Participants) | 47 | 39 | 44 | 44 | 43 | 38 | 43 | 46
  ENV peptide pool Mos2 at W 26 | 72.3 [57.36 to 84.38] | 41.0 [25.57 to 57.9] | 34.1 [20.49 to 49.92] | 72.7 [57.21 to 85.04] | 72.1 [56.33 to 84.67] | 71.1 [54.1 to 84.58] | 53.5 [37.65 to 68.82] | 2.2 [0.06 to 11.53]
  ENV peptide pool Mos2 at W 50: number analyzed (Participants) | 39 | 35 | 40 | 38 | 33 | 36 | 30 | 36
  ENV peptide pool Mos2 at W 50 | 84.6 [69.47 to 94.14] | 62.9 [44.92 to 78.53] | 37.5 [22.73 to 54.2] | 92.1 [78.62 to 98.34] | 87.9 [71.8 to 96.6] | 80.6 [63.98 to 91.81] | 60.0 [40.6 to 77.34] | 2.8 [0.07 to 14.53]
  ENV peptide pool potential T-cell epitopes(PTE)W26: number analyzed (Participants) | 47 | 39 | 44 | 44 | 43 | 38 | 43 | 46
  ENV peptide pool potential T-cell epitopes(PTE)W26 | 76.6 [61.97 to 87.7] | 59.0 [42.1 to 74.43] | 61.4 [45.5 to 75.64] | 72.7 [57.21 to 85.04] | 93.0 [80.94 to 98.54] | 81.6 [65.67 to 92.26] | 69.8 [53.87 to 82.82] | 2.2 [0.06 to 11.53]
  ENV peptide pool PTE at W 50: number analyzed (Participants) | 41 | 38 | 41 | 39 | 34 | 37 | 34 | 38
  ENV peptide pool PTE at W 50 | 80.5 [65.13 to 91.18] | 63.2 [45.99 to 78.19] | 58.5 [42.11 to 73.68] | 79.5 [63.54 to 90.7] | 88.2 [72.55 to 96.7] | 81.1 [64.84 to 92.04] | 67.6 [49.47 to 82.61] | 0 [0 to 9.25]
  ENV peptide pool PTE at W 78: number analyzed (Participants) | 41 | 36 | 0 | 0 | 0 | 0 | 0 | 0
  ENV peptide pool PTE at W 78 | 61.0 [44.5 to 75.8] | 50.0 [32.92 to 67.08] |  |  |  |  |  |
  ENV peptide pool PTE at W 96: number analyzed (Participants) | 39 | 32 | 25 | 22 | 23 | 24 | 21 | 0
  ENV peptide pool PTE at W 96 | 64.1 [47.18 to 78.8] | 40.6 [23.7 to 59.36] | 40.0 [21.13 to 61.33] | 50.0 [28.22 to 71.78] | 73.9 [51.59 to 89.77] | 62.5 [40.59 to 81.2] | 47.6 [25.71 to 70.22] |
  Gag peptide pool Mos1 at W 26: number analyzed (Participants) | 47 | 39 | 44 | 44 | 43 | 38 | 43 | 46
  Gag peptide pool Mos1 at W 26 | 44.7 [30.17 to 59.88] | 38.5 [23.36 to 55.38] | 36.4 [22.41 to 52.23] | 54.5 [38.85 to 69.61] | 55.8 [39.88 to 70.92] | 50.0 [33.38 to 66.62] | 34.9 [21.01 to 50.93] | 0 [0 to 7.71]
  Gag peptide pool Mos1 at W 50: number analyzed (Participants) | 41 | 38 | 41 | 39 | 34 | 36 | 34 | 38
  Gag peptide pool Mos1 at W 50 | 46.3 [30.66 to 62.58] | 47.4 [30.98 to 64.18] | 24.4 [12.36 to 40.3] | 61.5 [44.62 to 76.64] | 73.5 [55.64 to 87.12] | 61.1 [43.46 to 76.86] | 23.5 [10.75 to 41.17] | 2.6 [0.07 to 13.81]
  Gag peptide pool Mos2 at W 26: number analyzed (Participants) | 47 | 39 | 44 | 44 | 43 | 38 | 43 | 46
  Gag peptide pool Mos2 at W 26 | 48.9 [34.08 to 63.94] | 35.9 [21.2 to 52.82] | 43.2 [28.35 to 58.97] | 56.8 [41.03 to 71.65] | 55.8 [39.88 to 70.92] | 68.4 [51.35 to 82.5] | 39.5 [24.98 to 55.59] | 2.2 [0.06 to 11.53]
  Gag peptide pool Mos2 at W 50: number analyzed (Participants) | 39 | 34 | 40 | 38 | 33 | 36 | 30 | 35
  Gag peptide pool Mos2 at W 50 | 59.0 [42.1 to 74.43] | 47.1 [29.78 to 64.87] | 35.0 [20.63 to 51.68] | 71.1 [54.1 to 84.58] | 78.8 [61.09 to 91.02] | 66.7 [49.03 to 81.44] | 43.3 [25.46 to 62.57] | 0 [0 to 10]
  Gag peptide pool PTE at W 26: number analyzed (Participants) | 47 | 39 | 44 | 44 | 43 | 38 | 43 | 46
  Gag peptide pool PTE at W 26 | 38.3 [24.51 to 53.62] | 30.8 [17.02 to 47.57] | 38.6 [24.36 to 54.5] | 47.7 [32.46 to 63.31] | 55.8 [39.88 to 70.92] | 50.0 [33.38 to 66.62] | 30.2 [17.18 to 46.13] | 0 [0 to 7.71]
  Gag peptide pool PTE at W 50: number analyzed (Participants) | 39 | 36 | 41 | 38 | 34 | 36 | 32 | 36
  Gag peptide pool PTE at W 50 | 43.6 [27.81 to 60.38] | 47.2 [30.41 to 64.51] | 34.1 [20.08 to 50.59] | 50.0 [33.38 to 66.62] | 64.7 [46.49 to 80.25] | 63.9 [46.22 to 79.18] | 21.9 [9.28 to 39.97] | 5.6 [0.68 to 18.66]
  Gag peptide pool PTE at W 78: number analyzed (Participants) | 41 | 36 | 0 | 0 | 0 | 0 | 0 | 0
  Gag peptide pool PTE at W 78 | 29.3 [16.13 to 45.54] | 33.3 [18.56 to 50.97] |  |  |  |  |  |
  Gag peptide pool PTE at W 96: number analyzed (Participants) | 39 | 32 | 25 | 22 | 23 | 24 | 21 | 0
  Gag peptide pool PTE at W 96 | 20.5 [9.3 to 36.46] | 25.0 [11.46 to 43.4] | 20.0 [6.83 to 40.7] | 27.3 [10.73 to 50.22] | 30.4 [13.21 to 52.92] | 33.3 [15.63 to 55.32] | 23.8 [8.22 to 47.17] |
  Pol peptide pool Mos1 at W 26: number analyzed (Participants) | 47 | 39 | 44 | 44 | 43 | 38 | 43 | 46
  Pol peptide pool Mos1 at W 26 | 80.9 [66.74 to 90.85] | 53.8 [37.18 to 69.91] | 56.8 [41.03 to 71.65] | 70.5 [54.8 to 83.24] | 81.4 [66.6 to 91.61] | 89.5 [75.2 to 97.06] | 58.1 [42.13 to 72.99] | 4.3 [0.53 to 14.84]
  Pol peptide pool Mos1 at W 50: number analyzed (Participants) | 40 | 36 | 41 | 38 | 34 | 36 | 33 | 38
  Pol peptide pool Mos1 at W 50 | 72.5 [56.11 to 85.4] | 55.6 [38.1 to 72.06] | 65.9 [49.41 to 79.92] | 76.3 [59.76 to 88.56] | 85.3 [68.94 to 95.05] | 91.7 [77.53 to 98.25] | 39.4 [22.91 to 57.86] | 2.6 [0.07 to 13.81]
  Pol peptide pool Mos2 at W 26: number analyzed (Participants) | 47 | 39 | 44 | 44 | 43 | 38 | 43 | 46
  Pol peptide pool Mos2 at W 26 | 85.1 [71.69 to 93.8] | 76.9 [60.67 to 88.87] | 68.2 [52.42 to 81.39] | 79.5 [64.7 to 90.2] | 86.0 [72.07 to 94.7] | 94.7 [82.25 to 99.36] | 69.8 [53.87 to 82.82] | 0 [0 to 7.71]
  Pol peptide pool Mos2 at W 50: number analyzed (Participants) | 39 | 34 | 39 | 38 | 33 | 36 | 29 | 35
  Pol peptide pool Mos2 at W 50 | 84.6 [69.47 to 94.14] | 70.6 [52.52 to 84.9] | 79.5 [63.54 to 90.7] | 92.1 [78.62 to 98.34] | 97.0 [84.24 to 99.92] | 100.0 [90.26 to 100] | 55.2 [35.69 to 73.55] | 0 [0 to 10]
  Pol peptide pool PTE at W 26: number analyzed (Participants) | 47 | 39 | 44 | 44 | 43 | 38 | 43 | 46
  Pol peptide pool PTE at W 26 | 83.0 [69.19 to 92.35] | 56.4 [39.62 to 72.19] | 61.4 [45.5 to 75.64] | 68.2 [52.42 to 81.39] | 86.0 [72.07 to 94.7] | 92.1 [78.62 to 98.34] | 67.4 [51.46 to 80.92] | 0 [0 to 7.71]
  Pol peptide pool PTE at W 50: number analyzed (Participants) | 39 | 35 | 41 | 38 | 33 | 36 | 32 | 36
  Pol peptide pool PTE at W 50 | 82.1 [66.47 to 92.46] | 54.3 [36.65 to 71.17] | 73.2 [57.06 to 85.78] | 86.8 [71.91 to 95.59] | 90.9 [75.67 to 98.08] | 94.4 [81.34 to 99.32] | 53.1 [34.74 to 70.91] | 0 [0 to 9.74]
  Pol peptide pool PTE at W 78: number analyzed (Participants) | 41 | 36 | 0 | 0 | 0 | 0 | 0 | 0
  Pol peptide pool PTE at W 78 | 78.0 [62.39 to 89.44] | 52.8 [35.49 to 69.59] |  |  |  |  |  |
  Pol peptide pool PTE at W 96: number analyzed (Participants) | 39 | 32 | 25 | 22 | 23 | 24 | 21 | 0
  Pol peptide pool PTE at W 96 | 71.8 [55.13 to 85] | 40.6 [23.7 to 59.36] | 60.0 [38.67 to 78.87] | 36.4 [17.2 to 59.34] | 56.5 [34.49 to 76.81] | 62.5 [40.59 to 81.2] | 33.3 [14.59 to 56.97] |

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were reported up to Week 336 for Group 1 and 2 and up to Week 96 for the other groups (Group 3, Group 4, Group 5, Group 6, Group 7, Group 8). Other adverse events (AEs) were reported for the main study only period up to Week 96 for all the group
Description: The full analysis set (FAS) included all randomized participants with at least one study vaccine administration documented regardless of the occurrence of protocol deviations. Participants in Group 1 and 2 who received all 4 vaccinations in main study continued in long-term extension phase after Week 96 up to Week 336.
Arm/Group | Group 1: Ad26/Ad26 + gp140 High Dose (HD) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) | Group 3: Ad26/Ad26 | Group 4: Ad26/MVA + gp140 HD | Group 5: Ad26/ MVA + gp140 LD | Group 6: Ad26/MVA | Group 7: Ad26/ gp140 HD | Group 8: Placebo/ Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49 | 0/49 | 0/48 | 0/49 | 0/49 | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 8/50 | 3/49 | 3/49 | 4/48 | 4/49 | 5/49 | 2/50 | 5/49
Other Adverse Events (participants affected / at risk) | 40/50 | 36/49 | 42/49 | 42/48 | 34/49 | 41/49 | 43/50 | 38/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ad26/Ad26 + gp140 High Dose (HD) (N=50) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) (N=49) | Group 3: Ad26/Ad26 (N=49) | Group 4: Ad26/MVA + gp140 HD (N=48) | Group 5: Ad26/ MVA + gp140 LD (N=49) | Group 6: Ad26/MVA (N=49) | Group 7: Ad26/ gp140 HD (N=50) | Group 8: Placebo/ Placebo (N=49)
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Local Swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corona Virus Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hiv Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis Bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tubo-Ovarian Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stab Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Blighted Ovum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Complication of Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foetal Death (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal Disorder (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adjustment Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Generalised Anxiety Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Miscarriage of Partner (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy of Partner (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ad26/Ad26 + gp140 High Dose (HD) (N=50) | Group 2: Ad26/Ad26 + gp140 Low Dose (LD) (N=49) | Group 3: Ad26/Ad26 (N=49) | Group 4: Ad26/MVA + gp140 HD (N=48) | Group 5: Ad26/ MVA + gp140 LD (N=49) | Group 6: Ad26/MVA (N=49) | Group 7: Ad26/ gp140 HD (N=50) | Group 8: Placebo/ Placebo (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 1 | 2 | 2 | 4 | 1
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bundle Branch Block Right (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Conduction Disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deafness Unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Thyroid Mass (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Eye Swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid Pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ocular Discomfort (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 2 | 2 | 3 | 0 | 4 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Lip Blister (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tongue Dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth Impacted (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Adverse Drug Reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chest Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Feeling Cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling Hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 4
Injection Site Bruising (General disorders) | 1 | 2 | 2 | 0 | 5 | 2 | 2 | 0
Injection Site Haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Hypersensitivity (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Pain (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 2 | 1
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food Allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute Hiv Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Amoebiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ascariasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial Vaginosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Body Tinea (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Candida Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chlamydial Infection (Infections and infestations) | 1 | 0 | 2 | 2 | 1 | 1 | 3 | 2
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis Infected (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Genital Herpes Simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Gonorrhoea (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Herpes Simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hookworm Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 4 | 3 | 5 | 5 | 5 | 1 | 6 | 5
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Malaria (Infections and infestations) | 2 | 2 | 3 | 1 | 1 | 3 | 2 | 2
Oophoritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis Externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parasitic Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 3
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pulpitis Dental (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pyuria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash Pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 2 | 2 | 1 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syphilis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinea Versicolour (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tooth Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trichomoniasis (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Typhoid Fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 6 | 2 | 6 | 5 | 7 | 6 | 9
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urethritis Chlamydial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 2 | 5 | 5 | 3 | 3 | 1 | 0
Urogenital Trichomoniasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral Infection (Infections and infestations) | 2 | 1 | 3 | 1 | 0 | 3 | 3 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 3 | 2 | 1 | 1
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vulvovaginitis Trichomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural Dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural Headache (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Stress Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 6 | 3 | 2 | 2 | 4 | 3 | 3 | 1
Aspartate Aminotransferase Increased (Investigations) | 4 | 1 | 4 | 1 | 2 | 3 | 3 | 2
Blood Creatine Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Creatinine Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 3 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Pressure Diastolic Increased (Investigations) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Blood Pressure Systolic (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Pressure Systolic Increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2
Blood Urine Present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT Prolonged (Investigations) | 2 | 1 | 3 | 3 | 0 | 4 | 2 | 2
Eosinophil Percentage Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin Decreased (Investigations) | 1 | 2 | 4 | 4 | 0 | 3 | 2 | 0
Neutrophil Count Decreased (Investigations) | 1 | 1 | 2 | 0 | 1 | 3 | 1 | 1
Platelet Count Decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Protein Urine (Investigations) | 2 | 0 | 0 | 0 | 2 | 2 | 1 | 3
Red Blood Cells Urine (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White Blood Cells Urine (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 4 | 1 | 2 | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Burning Sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 1
Dizziness Exertional (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dizziness Postural (Nervous system disorders) | 1 | 1 | 3 | 1 | 1 | 2 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 4 | 5 | 3 | 1 | 4 | 2 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Affective Disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Libido Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 2 | 3 | 0 | 2 | 1 | 2
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 4 | 4 | 2 | 3 | 1 | 4 | 6 | 4
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast Tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Genital Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital Rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital Ulceration (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Premenstrual Syndrome (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 4 | 2 | 2 | 4 | 1
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 3 | 2 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pregnancy of Partner (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Systolic Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT02315703/Prot_002.pdf
  • Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT02315703/SAP_003.pdf